

A single-centre Phase1b study to assess the safety, tolerability, pharmacokinetic profile, and antimalarial activity of single doses of coadministered artefenomel (OZ439) and piperaquine phosphate (PQP) against earl plasmodium falciparum blood stage infection in healthy adult volunteers

Protocol Identifying Number: QP17C19

Principal Investigator: Prof. James McCarthy

Study Sponsor Medicines for Malaria Venture

Local Sponsor: Clinical Network Services

Version Number: Protocol 4.0

27 August 2018

#### CONFIDENTIALITY STATEMENT

This document contains information that privileged or confidentialAs such, it may not be disclosed unless specific prior permission is granted in writingledicines for Malaria Venture or such disclosure is required by federal or other laws or regusalTersons to whom any of this information is to be disclosed multist be informed that information is confidentialThese restrictions on disclosure will apply equally to all future information supplied, which is indicated as privileged or confidential

| CONTENT | S | |
|---|---|---|
| LIST OF AE | BBREVIATION S | 1 |
| STATEMENT | COF COMPLIANCE | 4 |
| PROTOCOL | SUMMARY | 6 |
| | C OF STUDY D ESIGN | |
| | ROLES | |
| | ODUCTION: BACKGR OUND INFORMATION AND SCIENTIFIC RATIO | |
| 18 | | |
| | BACKGROUND INFORMATION | |
| | RATIONALE | |
| 2.3 | POTENTIAL RISKS AND BENEFITS | |
| 2.3.1 | KNOWN POTENTIAL RISKS | |
| 2.3.2 | KNOWN POTENTIAL BENEFITS | |
| | ECTIVES AND PURPOSE | |
| | DY DESIGN AND ENDPOINTS | |
| | DESCRIPTION OF THE SUDY DESIGN | |
| | STUDY ENDPOINTS | |
| 4.2.1 | PRIMARY ENDPOINT | |
| 4.2.2 | SECONDARY ENDPOINTS | |
| 4.2.3 | EXPLORATORY ENDPOINTS | |
| | DY ENROLLMENT AND WITHDRAWAL | |
| | Subject Inclusion Criteria | |
| | Subject Exclusion Criteria | |
| | Contraception | |
| | Strategies for Recruitment and Retention | |
| | Subject Withdrawal or termination | |
| 5.5.1 | Reasons for Withdrawal or Termination | |
| 5.5.2 | Handling of Subject Withdrawals or termination | |
| | Premature Termination or Suspension of Study | |
| | DY AGENT | |
| | STUDY AGENT(S) AND CONTROLDESCRIPTION | |
| 6.1.1 | ACQUISITION | |
| 6.1.2<br>6.1.3 | FORMULATION, APPEARANCE, PACKAGING, AND LABELING PRODUCT STORAGE AND STABILITY | |
| 6.1.4<br>6.1.5 | PREPARATIONDOSING AND ADMINISTRATION | |
| 6.1.5 | ROUTE OF ADMINISTRATION | |
| 6.1.7 | STARTING DOSE AND DOSE ESCALATION SCHEDULE | |
| 6.1.8 | DOSE ADJUSTMENTS/MODFICATIONS/DELAYS | |
| 6.1.9 | Duration of Therapy | |
| 6.1.10 | Tracking of Dose | |
| | Study agent Accountability Procedures | |
| | OY PROCEDURES AND SCHEDULE | |
| | STUDY PROCEDURES/EVAUATIONS | |
| 7.1.1 | STUDY SPECIFIC PROCBURES | |
| 7.1.2 | STANDARD OF CARE STIDY PROCEDURES | |

| 7.2 | LABORATORY PROCEDURES/EVALUATIONS | 51 |
|--------|--------------------------------------------------------|-------|
| 7.2.1 | CLINICAL LABORATORY EVALUATIONS | 51 |
| 7.2.2 | Other Assays or Procedures | |
| 7.2.3 | SPECIMEN PREPARATION HANDLING, AND STORAGE | 56 |
| 7.2.4 | SPECIMEN SHIPMENT | 56 |
| 7.3 | STUDY SCHEDULE | 56 |
| 7.3.1 | SCREENING | 56 |
| 7.3.2 | ELIGIBILITY CONFIRMATION VISIT | 58 |
| 7.3.3 | FOLLOW-UP | 59 |
| 7.3.4 | END OF STUDY VISIT (EOS) | 63 |
| 7.3.5 | EARLY TERMINATION VI SIT | 64 |
| 7.3.6 | UNSCHEDULED VISIT | 64 |
| 7.3.7 | SCHEDULE OF EVENTS TABLE | 64 |
| 7.4 | JUSTIFICATION FOR SENSITIVE PROCEDURES | 69 |
| 7.5 | CONCOMITANT MEDICATIONS, TREATMENTS, ANDPROCEDURES | 69 |
| 7.5.1 | PRECAUTIONARY MEDICATIONS, TREATMENTS, AND PROCE 69 | DURES |
| 7.6 | PROHIBITED MEDICATIONS, TREATMENTS, ANDPROCEDURES | 69 |
| 7.7 | PROPHYLACTIC MEDICATIONS, TREATMENTS, AND PROCEDURES | 70 |
| 7.8 | RESCUE MEDICATIONS, TREATMENTS, AND PROCEDURES | 70 |
| 7.9 | SUBJECT ACCESS TO SUTDY AGENT AT STUDY CLOSURE | 70 |
| 8 ASS | SESSMENT OF SAFETY | 7.0 |
| 8.1 | SPECIFICATION OF SAETY PARAMETERS | |
| 8.1.1 | DEFINITION OF AES (AE) | 7.0 |
| 8.1.2 | DEFINITION OF SERIOUS AES (SAE) | 7.2 |
| 8.1.3 | DEFINITION OF AES OF SPECIAL INTEREST (AESI) | 7.3 |
| 8.2 | CLASSIFICATION OF ANAE | 74 |
| 8.2.1 | SEVERITY OF EVENT | 74 |
| 8.2.2 | RELATIONSHIP TO STUDY AGENT | 75 |
| 8.2.3 | EXPECTEDNESS | 76 |
| 8.3 | TIME PERIOD AND FREQUENCYFOR EVENT ASSESSMENTAND FOLLO | )W-UP |
| 8.4 | REPORTING PROCEDURES | 77 |
| 8.4.1 | AE REPORTING | 77 |
| 8.4.2 | SERIOUS AE REPORTING | 79 |
| 8.4.3 | UNANTICIPATED PROBLEM REPORTING | 80 |
| 8.4.4 | AES OF SPECIAL INTEREST (AESI) | 80 |
| 8.4.5 | REPORTING OF PREGNARY | |
| 8.5 | STUDY HALTING RULES | 80 |
| 8.6 | SAFETY OVERSIGHT | 81 |
| 9 CLII | NI CAL MONITORING | 81 |
| | TISTICAL CONSIDER ATIONS | |
| 10.1 | STATISTICAL ANALYSIS PLAN | _ |
| 10.2 | ANALYSIS DATASETS | 82 |
| 10.3 | DESCRIPTION OF STATISTICAL METHODS | 82 |
| 10.3.1 | GENERAL APPROACH | 82 |
| 10.3.2 | ANALYSIS OF THE PRIMARY EFFICACY ENDPOINT(S) | 83 |

| 10.3.3 | ANALYSIS OF THE SECONDARY ENDPOINT(S) | 83 |
|---|---|---|
| 10.3.4 | SAFETY ANALYSES | |
| 10.3.5 | ADHERENCE AND RETENTION ANALYSES | |
| 10.3.6 BASEL | INE DESCRIPTIVE STATISTICS | |
| 10.3.7 | PLANNED INTERIM ANALYSES | 85 |
| 10.3.8 | ADDITIONAL SUB-GROUP ANALYSES | 85 |
| 10.3.9 | MULTIPLE COMPARISONMULTIPLICITY | 86 |
| 10.3.10 TABU | LATION OF INDIVIDUAL RESPONSE DATA | 86 |
| 10.3.11 EXPL | ORATORYANALYSES | 86 |
| 10.4 SAMPI | LE SIZE | 86 |
| 10.5 MEASU | URES TO MINIMIZE BIAS | |
| 10.5.1 | ENROLLMENT/ RANDOMIZATION/ MASKING PROCEDU | |
| 10.5.2 | EVALUATION OF SUCCESS OF BLINDING | 86 |
| 10.5.3 | BREAKING THE STUDY BLIND/SUBJECT CODE | 86 |
| 11 SOURCE DO | OCUMENTS AND ACCESS TO SOURCE DATA/DOCUMENT | s87 |
| 12 QUALITY AS | SSURANCE AN D QUALITY CONTROL | 87 |
| 13 ETHICS/PR | OTECTION OF HUMAN SUBJECTS | 87 |
| | AL STANDARD | |
| | AL REVIEW | |
| 13.3 INFOR | MED CONSENT PRŒESS | |
| 13.3.1 | CONSENT/ASSENT AND OTHER INFORMATIONAL | |
| PROVIDED TO | OSUBJECTS | |
| 13.3.2 | CONSENT PROCEDURES NO DOCUMENTATION | |
| | ECT AND DATA CONFIDENTIALITY | |
| 13.4.1 | RESEARCH USE OF STORD HUMAN SAMPLES, SÆCIM<br>91 | ENS OR DATA |
| 13.5 FUTUF | RE USE OF STOREDSPECIMENS | 91 |
| 14 DATA HAND | DLING AND RE CORD KEEPING | 92 |
| 14.1 DATA | COLLECTION AND MANAGEMENT RESPONSIBLITIES | 92 |
| 14.2 STUDY | Y RECORDS RETENTON | 92 |
| 14.3 PROT | OCOL DEVIATIONS | 93 |
| 14.4 PUBLI | CATION AND DATA SHARING POLICY | 93 |
| 15 STUDY ADM | MINISTRATION | 95 |
| | Y LEADERSHIP | |
| 15.2 LIABIL | .ITY/INDEMNITY/ INSURANCE | 95 |
| 16 CONFLICT | OF INTEREST POLICY | 95 |
| 17 LITERATUR | RE REFERENCE S | 95 |

| LIST OF ABBREVIAT | ION S |
|---|---|
| ACPR | Adjusted Adequate Clinical and Parasitological Response |
| ACT | Artemisinin Combination Therapy |
| AE | AE |
| AESI | AE of Special Interest |
| ALT | Alanine Aminotransferase |
| ANZCTR | Australia New Zealand Clinical Trial Registry |
| anti-HBc Ab | Anti-Hepatitis B Core Antibodies |
| anti-HCV | Anti-Hepatitis C Virus |
| anti-HIV1 | Anti-Human Immunodeficiency Virus 1 |
| anti-HIV2 | Anti-HumanImmunodeficiency Virus 2 |
| AST | Aspartate Aminotransferase |
| AUC | Area Under the Curve |
| AUC <sub>inf</sub> | AUC Curve to Infinite Time |
| AUC <sub>last</sub> | AUC Curve to Last Quantifiable Concentration |
| BDI | Beck Depression Index |
| Blood Service | Australian Red Cross Blood Service |
| CRP | C-Reactive Protein |
| C <sub>max</sub> | Maximum Plasma Concentration |
| CNS | Clinical Network Services |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria fokEs |
| eCRF | Electronic Case Report Form |
| ECG | Electrocardiogram |
| EC <sub>50</sub> | Half maximal effective concentration |
| EOS | End of Study |
| E <sub>max</sub> | Maximum effective concentration |
| FDA | Food and Drug Administration |
| FSH | Follicle-Stimulating Hormone |
| FQ | Ferroquine |
| G6PD | Glucose6-Phosphate Dehydrogenase |
| GCP | Good Clinical Practice |
| GI | Gastrointestinal |
| GMP | Good Manufacturing Practice |
| GPDI | General Pharmacodynamic Interaction |
| HAV | Hepatitis A Virus |
| HBs Ag | Hepatitis B surface antigen |
| HCV | Hepatitis C Virus |
| HEV | Hepatitis E Virus |
| HDL | High Density Lipoprotein |
| HIV | Human Immunodeficiency Virus |
| HPLC | High-Performance Liquid Cromatograph System |
| HREC | Human Research Ethics Committee |

| IB | Investigatos Brochure |
|---|---|
| IBSM | Induced Blood Stage Malaria |
| ICH | International Conference on Harmonization |
| IMM | Independent Medical Monitor |
| IMP | Investigational Medicinal Product |
| IV | Intravenous |
| LC MS | Liquid ChromatographyMassSpectrometry |
| LFT | Liver Function Test |
| LLOQ | Lower Limit of Quantification |
| MAP | Modelling Analysis Plan |
| MCB | Master Cell Bank |
| MedDRA | Medical Dictionary for Regulator Activities |
| MFA | Membrane Feeding Assay |
| MIC | Minimum Inhibitory Concentration |
| MMV | Medicines for Malaria Venture |
| MPC | Minimal Parasiticidal Oncentration |
| NHMRC | National Health and Medical Research Council |
| NLME | Non-linear mixed effect |
| NTF | Note To File |
| OZ439 | Artefenomel |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| PK/PD | Pharmacokinetic/Pharmacodynamic |
| PQP | Piperaquine Phosphate |
| PRR | Parasite Reduction Ratio |
| Pt <sub>½</sub> | Parasite clearance hailfe |
| QIMR Berghofer | Queensland Institute of Medical Research Berghofer |
| qPCR | Quantitative Polymerase Chain Reaction |
| qRT-PCR | QuantitativeReverse Transcription Polymerase Chain Reaction |
| QTc | Corrected QT |
| RBC | Red Blood Cell |
| Rh | Rhesus Antibody |
| SAE | SeriousAE |
| SAP | Statistical Analysis Plan |
| SDRT | Safetyand DataReviewTeam |
| SERC | Single Exposure Radical Cure |
| SOP | Standard Operating Procedures |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| t <sub>1/2</sub> | Terminal HalfLife |
| TEAE | TreatmentEmergentAE |
| TGA | Therapeutic Goods Administration |
| T <sub>max</sub> | Time taken to reach |
| TPGS | α-tocopherol polyethylene glycol 1000 succinate |

| TPP | Target Product Profile |
|-------|---------------------------------|
| ULN | Upper Limit of Normal |
| WHO | World Health Organization |
| WOCBP | Women of Childbearing Potential |

# STATEMENT OF COMPLIA NCE

#### **Investigator declaration**

I have read the protocol and agree that it contains all necessary details for carrying out the study as described. I will conduct this otocol as outlined herein and will make a reasonable effort to complete the study within the time designated.

I agree to personally conduct or supervise the described.

The study will be conducted in accordance with the following:

- World Medical Association Declaration of Helsinki- Ethical Principles for Medical Research Involving Huma Bubjects (Fortaleza, Brazil 2013)
- NHMRC National Statement on Ethical Conduct in Human Research, (2007 ted May 2015).
- Note for Guidance on Good Clinical Practi(GCP)

   – Annotated with Therapeutic Goods
   Administration(TGA) Comments (CPMP/ICH/135/95), as adopted by Atbstralian TGA
   (July 2000)
- Current ethics approved Clinical Trial Protocol

I agree to inform alsubjects that the study drusgarebeing used or investigational purposes and I will ensure that the requirements related to obtaining informed consent are in accordance with International Council of Harmonisation (CH) Guidelines for GCP Section 4.8 and local requirements.

I agree to report that occur in the course of the Sponsor in accordance with ICH Guidelines for GCP ection 4.11 and local requirements.

I have read and understand the information inhomestigators Brochures, including the potential risks and side effects the studydrugs.

I agree to promptly report to the uman Research thics Committee (REC) all changes in the research activity and all unanticipated problems involving risturbjects. I will not make any changes to the conduct of the study with the REC and Sponsor approval, except when necessary to eliminate apparent immediate harmstopjects.

I agree to maintain adequate and accurate records and make those records available in accordance with ICH Guidelines for GCE ection 4.11 and local requirement

I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed about their obligations in meeting the above commitments.

I understand that the udy may be terminated or enrolment suspended at anybyinthe Sponsor, with or without cause, or by me if it becomes necessary to protect the best interestuble by:

| | Date: |
|--------------------------------------------|-------|
| Professor James McCarth rincipal Investiga | ator |

# Signatories

The undersigned parties agree that the protocol was written in accordance with the World Medical Association Declaration of Helsinki Ethical Principles for Medical Research Involving Human Subjects (Fortaleza, Brazil 2013), the HMRC National Statement on Ethical Conduct in Human Research (2007, updated May 2015) depend the Note or Guidance on Good Clinical Practice Annotated with TGA Comments (CPMP/ICH/135/95), as adopted by the Eralian Therapeutic Goods Administration July 2000).

| Name | Signature | Date |
|-------------------------------------------|-----------|------|
| Protocol Writer: | | |
| Dr Rebecca WebsterPhD | | |
| Clinical Trials Project Manager | | |
| QIMR Berghofer Medical Research Institute | | |

This clinical trial protocol has been reviewed and approved by the Sponsor.

| Name | Signature | Date |
|-------------------------------|-----------|------|
| SponsorMedical Director. | | |
| Stephan Chalon MD, PhD | | |
| Medicines for Malaria Venture | | |
| Sponsor Project Director: | | |
| Jörg Möhrle PhD | | |
| Medicines for Malaria Venture | | |

# PROTOCOL SUMMARY

| Title: | A single-centre Phase b1 study to assess the safety, tolerabil |
|---|---|
| | pharmacokinetic profile, and antimalarial activity of single doses of |
| | administeredartefenomel (OZ439) and piperaquine phosphate (P |
| | against earlyPlasmodiunfalciparum blood stage infection in health |

adult volunteers.

# Study Description:

This is a singlecentre, open label, adaptive study using the P. falciparum induced blood stage malar (LBSM) inoculum as a mode to character is the pharmacodynamic (PD) activity of combined single dose administration of OZ439 and PQP

The study will be conducted in a maximum of three cohorts (up subjects per cohort) using up to 4 different dosses Z439 and PQP in each cohort Subjects will be malaria naïve healthy males or females between 18-55 years old, who meet all of the inclusion criteria anothe of the exclusion criteria.

The first cohort will be composed 4 groups of 2 subjects each Subjects will be randomised into one of dosegroups and administered single of doses of OZ439 and PQP in combination to each of the groups in this cohort as show in Table 1.

Table 1 OZ439 and PQP Cohort 1 Dose

| Drug | Dose group | | | |
|-----------|------------|-----|-----|-----|
| | 1A | 1B | 1C | 1D |
| OZ439(mg) | 200 | 200 | 400 | 400 |
| PQP (mg) | 480 | 640 | 480 | 640 |

The data captured from this first cohort will be used to determine relationship between OZ439 and PQP concentrations and parasit levels Based onsafety and tolerability data up to Day42±2 and pharmacokinetic/pharmacodynamic (PK/PD) alysis outcomes (based PD data up to Day42±2 and PK data up to Day5±2), the dos(s) for the subsequent ohortwill be determined.

After review of the PK/PD and safety data from Cohort 1 by Statety and DataReviewTeam (SDRT) it was determine that, the second cohor will be composed of 2 dose groups 4 subjects each Subjects will be randomised into one of dose groups and administered single oral do of OZ439 and PQP in combination the combined dose of Z439 and PQP will be different for each group in this cohort as shown in Table 2.

Table 2 OZ439 and PQP Cohort2 Dose

| Drug | Dose group | |
|-----------|------------|-----|
| | 2A | 2B |
| OZ439(mg) | 800 | 200 |
| PQP (mg) | 960 | 320 |

A similar analysis will be done at the end of cohort 2 combining control and 2 data to decide the doseto be tested in cohort 3. his will be decided by the funding sponsor and the incipal Investigator following review of the data by the DRT and scientific evaluation.

The doses used in cohorts will not exceed the maximum acceptal doses predefined for this study (800 mg for OZ439 and 1440 mg for as determined in previous safety, pilot efficacy and phase 2 studies.

Each subject will be inoculated on Day 0 with approximately 2,800 viparasites of P. falciparum-infected human erythrocytes administer intravenously. Subjects will be blowed updaily via phone calbr text messagen Days 1 to 3 postnoculation to solicit any AEs.

Subjects will then come to the clinical unit one daily from Day 4 until presence of asexual parasites is established by quantitative polyr chain reaction (qPCR) targeting the 18S rRNA gene (referred to asmalaria 18S qPCR). Once qPCR comespositive and until OZ439 and PQP administration subjects will come to the clinical unit twicedaily, separated by approximately 12 hours, for clinical evaluation and to sampling.

Subjectswill be admitted to the linical unit for single dose administration of OZ439 and PQP days after malaria invalation or earlier if a subject has a malaria clinical score > 6r at Investigatos discretion Subjects will

be followed up as inpatients for at least 72 hours to ensure tolerance investigational treatments and clinical response, then if clinically well of an outpatient basis for safety and clearance of malaria parasites via

After discharge from the clinical unit subjects will be followed up regularly for safety assessments, PK sampling, clinierabilization, and malaria qPCR blood sampling unitary 42±2 (34 days after OZ439 an PQP administration All subjects will receive a standard course of ther with Riamet® (artemethelumefantrine) on Day 42±2, or earlier in the event of failure of clearancer recrudescence of parasitaemoia at Investigators discretiorbased on subject safety or guidance, the definitions for failure of parasite clearance and recrudescence are definitions.

- Failure of clearancedefinedasfailure to clear parasitaemia by least 10 fold at 72 hours postMP administration
- Recrudescencetefined as 5 000 blood stage parasites/mL and a
   2-fold parasitaemiancrease within 48 hours, re-occurrence f
   malaria symptoms with malaria clinical score >6)

The presence of gametocytes in subjects' blood will be determined by parasite lifecycle stage qRFCR or by the presence of stable low le parasitaemialf gametocytes are present the time of treatment wit Riamet® Primacin<sup>TM</sup> (primaquine) will also be administered as a single oral dose

AEs (AEs) will be monitored via telephone, within the clinical unit, a on outpatient review after malaria challenge inoculation and antima study drugs administration. Bloodraples for safety evaluation, malar monitoring, and red blood cell antibodies will be drawn at screening a baseline and at nominated times after malaria challenge.

# Objectives:

#### Primary:

The primary study objectives are:

- a. To charactese the PK/PD relationshipetweenOZ439 and PQF plasma concentrations and blood stage aseparatisitaemian healthy subjects following. falciparumIBSM infection.
- b. To evaluate the safety and tolerability of OZ439 and PQP whe administered as singledoses in healthysubjects following P. falciparum IBSM infection

# Secondary:

The secondary study objectives are:

- a. To describe the PK of OZ439 and PQP wheradministered as single doses in healthy volunteers under fasted conditions.
- To characterize the PD effect of-administered single doses OZ439 and PQP on clearance falciparumasexual blood stag parasites from the blood of healthy subjects in the IBSM mod

## Exploratory:

The exploratorystudy objectives are:

- a. To charactese specific cell subsets and immune signate associated with control of parasite burden and pathoger following first exposure to falciparum to identify specific cells immunomodulatory molecules and immune pathways to targe therapeuticintervention
- To investigate the role of RBC complement regulatory proteins anti-phosphatidylserine antibodies in malarial anaemia
- c. To investigate the association between serum comple activation, complement activating antibodies, and R complementegulatory protein expression

#### **Endpoints:**

### Primary:

Primary study endpoints:

- a. The PK/PD relationship between OZ439 and PQP pla concentrations and blood stage asexual parasitaemia wi determined by:
  - Effect of OZ439 on Emax and EC50 of PQP
  - Effect of PQP on Emax and EC50 of OZ439
- b. The incidence, severity and relationship to OZ439 and PQ observed and selfeportedAEs up to trial Day 422 after the co-administration of single doses of OZ439 and PQPhealthy subjects inoculated ith IBSM

# Secondary:

Secondary study endpoints:

- a. Estimation of OZ439 and PQP PK parameters trial Day 422 of single doses using nonempartmental methods: AUC068h, AUClast, AUC0inf, Cmax, tmax, t1/2, tlag, C168 CL/F, Vz/F and λinf.
- b. The effect of coadministered single oral doses of OZ439 and F on clearance of falciparumblood stage parasites from the blo of inoculated subjects as measured by qRPR trial Day 422. Parasite clearance will be assessed by the following paramet
  - Parasite clearance hailfe (Pt ½),
  - Parasite reduction ratio (PRR),
  - Percentage of subjects with recrudescence of parasital defined as 5 000 blood stage parasites/mL and a 2-fold increase within 48 hours, or -cecurrence of malarial symptoms with a malarial clinical score >6)

| | Exploratory: |
|---|---|
| | a. Identification of immune checkpoint molecules |
| | <ul> <li>b. The level of expression of complement regulators/teins (CD35,<br/>CD55 and CD59) and phosphatidylserine on RBC.</li> </ul> |
| | c. The level of <b>c</b> mplement activating antibodies and ar phosphatidylserine antibodies |
| Population: | A total of up to24 subjects will be enrolled in this studyp( to 3 cohorts of 8 subjects each). Subjects will be malaria naïve healthy male females aged between 1855 years old, who meet all of the inclusi criteria and none of the exclusion criteria |
| | In each cohort, if morthan, 2 discontinuations due to nonafety related reasons occur; additional subjects may be recruited to replace discontinued subjects on agreement with the study sponsor. |
| | Subjects eligible for inclusion of the study will be further invited participate in optional exploratory omponents that ill require additional blood samples to be taken at scheduled -timiets during the study Details regarding these optional study components will be provided separate Participant Information Sheet and subjects agreeing to part in these components with rovide specific written consent for this. Refuse to participate in the optional study components will not jeopardissubjects' participation in the main study. |
| Phase: | Phase 1b |
| Number of sites enrolling subjects: | The study is planned to be perform one investigational site: Q-Pharm Pty Ltd Level 5, 300C Herston Rd and Level 6, Block 8, Royal Brisbane and Women's Hospital Herston QLD 4006, Australia Additional sites in Australia may be added if necessary. |
| Description of study agents: | Malaria challenge agent: P. falciparum3D7 blood stage challenge agent |

The P. falciparum 3D7 master cell bank (MCB) was produced from blocollected from a donor with clinical manifestation of mala Each 3D7 inoculum dose will be prepared aseptically from a doubt of the P. falciparum 3D7 MCB. Each subject administered 3D7 will inoculated intravenously with a dose of approximately 2,800 viable P. falciparum 3D7-infected RBCsin 2 mL of saline for injection.

Investigational medicinal products:

#### OZ439

 $OZ439 + \alpha$ -tocopherol polyethylene glycol 1000 succinate (TPG granules for oral suspension, in 200 amgl400 mg dosages and provid with sucrose

#### **PQP**

Piperaquine phosphate (PQP), 160 tables.

Antimalarial rescue medications:

#### Artemether/lumefantrie

Riame® (20 mg artemether and 120 mg lumefantrine) will administered to all subjects beginning on approximately \$\mathbb{D}\alpha\bar{2}\$ (34 days after administration of OZ439 and PQR) rearlier in the event of failure of clearance recrudescence of parasitae miaat Investigators discretion based on subject safety course of treatment comprises 6 do of 4 tablets administered orally over a period of 60 hours (total cour 24 tablets). Each dose of tablets should be taken with food or drink in fat (e.g., milk).

#### Primaquine(if required)

Subjects may receivæsingleoral dose of Primacin<sup>™</sup> equivalent to 45 mg primaquine (6 tablets, each containing primaquine phosphate 13. equivalent to 7.5 mg of primaquine) to ensure complete clearanc gametocytes.

#### Artesunate (if required)

Treatment of subjects with intravenous sesunate will only occur in the event that subjects are unable to complete oral treatment wither (e.g. the subject is vomiting). Treatment with artesunate ould be done at the recommended dose regime f 2.4 mg/kg at approximately 0, 12, 24, hours and then daily for up to 7 days or until able to take oral drugs.

| Duration of Study | It is estimated that the clinical portion of the study will be completed approximately 10 months |
|---|---|
| Duration subject participation: | Approximately 25 months (74 days) for eachsubject including a screening period of up to 28 days, a period of observation follo inoculation of approximately8 days, and a followup period after administration of OZ439 and PQP3 days. |

# SCHEMATIC OF STUDY DESIGN



# OZ439 + PQP Combination



# KEY ROLES

| PrincipalInvestigator Prof. James McCarthy, MBBS Q-Pharm Pty Ltd (visiting Medical Officer) and QIMR Berghofer Medical Research Institute Level 5, 300C Herston Rd Herston QLD 4006, Australia Tel: +61(0)7 3845 3647 or +61 (0)7 3845 3636 Mobile: +61 4144204659 Email: j.mccarthy@uq.edu.au Co-Investigato/s Dr Paul Griffin MBBS FRACP FRCPA Q-Pharm Pty Ltd Level 5, 300C Herston Road Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au Dr Anand Odedra MBBS |
|---|
| QIMR Berghofer Medical Research Institute Level 5, 300C Herston Rd Herston QLD 4006, Australia Tel: +61(0)7 3845 3647 or +61 (0)7 3845 3636 Mobile: +61 4144204659 Email: j.mccarthy@uq.edu.au Co-Investigato/s Dr Paul Griffin MBBS FRACP FRCPA Q-Pharm Pty Ltd Level 5, 300C Herston Road Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Level 5, 300C Herston Rd Herston QLD 4006, Australia Tel: +61(0)7 3845 3647 or +61 (0)7 3845 3636 Mobile: +61 4144204659 Email: j.mccarthy@uq.edu.au Co-Investigato/s Dr Paul Griffin MBBS FRACP FRCPA Q-Pharm Pty Ltd Level 5, 300C Herston Road Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Herston QLD 4006, Australia Tel: +61(0)7 3845 3647 or +61 (0)7 3845 3636 Mobile: +61 4144204659 Email: j.mccarthy@uq.edu.au Co-Investigato/s Dr Paul Griffin MBBS FRACP FRCPA Q-Pharm Pty Ltd Level 5, 300C Herston Road Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Tel: +61(0)7 3845 3647 or +61 (0)7 3845 3636 Mobile: +61 4144204659 Email: j.mccarthy@uq.edu.au Co-Investigato/s Dr Paul Griffin MBBS FRACP FRCPA Q-Pharm Pty Ltd Level 5, 300C Herston Road Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Mobile: +61 4144204659 Email: j.mccarthy@uq.edu.au Co-Investigato/s Dr Paul Griffin MBBS FRACP FRCPA Q-Pharm Pty Ltd Level 5, 300C Herston Road Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Email: j.mccarthy@uq.edu.au Co-Investigato/s Dr Paul Griffin MBBS FRACP FRCPA Q-Pharm Pty Ltd Level 5, 300C Herston Road Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Co-Investigato/s Dr Paul Griffin MBBS FRACP FRCPA Q-Pharm Pty Ltd Level 5, 300C Herston Road Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Q-Pharm Pty Ltd Level 5, 300C Herston Road Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Level 5, 300C Herston Road Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Herston QLD 4006, Australia Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Tel: +61 (0)7 3845 3647 Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Fax: +61 (0)7 3845 3637 Email: paul.griffin@infectiousdiseasesqld.com.au |
| Email: paul.griffin@infectiousdiseasesqld.com.au |
| Dr Anand Odedra MBBS |
| Q-Pharm Pty Ltd (visiting Medical Officer) and |
| QIMR Berghofer Medical Research Institute |
| Level 5, 300C Herston Road |
| Herston QLD 4006, Australia |
| Tel: +61 (0)7 3845 3636 |
| Email: Anand.Odedra@qimrberghofer.edu.au |
| Dr Bridget BarbeiMBBS, DTM&H, MPH, FRACP, PhD |
| Q-Pharm Pty Ltd (visiting Medical Officer) and |
| QIMR Berghofer Medical Research Institute |
| Level 5, 300C Herston Road |
| Herston QLD 4006, Australia |
| Tel: +61 424737153 |
| Email: BridgetBarber@qimrberghofer.edu.au |
| Local Sponsor/s Clinical Network Services (CNS) Pty Ltd |
| Level 4, 88 Jephson St |
| Toowong QLD 4066, Australia |
| Tel: +61 (0)7 3719 6000 |
| Sponsor Medical Director Stephan Chalon, MD, PhD |
| Medicines for Malaria Venture |
| Route de Presois 20 |
| 1215 Geneva 15 |

| | Switzerland |
|---|---|
| | Email: chalons@mmv.org |
| Sponsor Project Director | Jörg Möhrle PhD |
| , | Medicines for Malaria Venture |
| | Route de PrésBois 20 |
| | 1215 Geneva 15 |
| | Switzerland |
| | Tel: +4122 555 0330 |
| Spangar Clinical Scientist | Email: moehrlej@mmv.org |
| Sponsor Clinical Scientist | Myriam El Gaaloul, PharmD |
| | Medicines for Malaria Venture |
| | Route de Presois 20<br>1215 Geneva 15 |
| | Switzerland |
| | Tel: +41 22 555 0377 |
| | Email: elgaaloulm@mmv.org |
| Medical Monitor | |
| Wedical Worldon | Dr. med. Michael Marx MD |
| | Medical Director |
| | ICON Clinical Research |
| | Internal Tel: 7123 1568 |
| | ExternalTel: +49 6103 904 1568 |
| | Mobile : (+49) 172 677 7401 |
| | Email: Michael.Marx@iconplc.com |
| MedicalMalaria Expert | Prof. Dennis Shanks |
| | Australian Army Malaria Institute |
| | Gallipoli Barracks |
| | Enoggera QLD 4051, Australia |
| | Tel: +61 (0)7 3332 4931 |
| | Email: Dennis.SHANKS@defence.gov.au |
| Institutional Ethics | QIMR Berghofer Medical Research Institute Human Rese |
| Committee | Ethics Committee (QIMR Berghofer HREC; EC00278) |
| | Locked Bag 2000, Royal Brisbane and Women's Hospital |
| | Brisbane QLD 4029, Australia |
| | Tel: +61 (0)7 3362 0117 |
| Sponsor Pharmacometrician | · |
| | Medicines for Malaria Venture |
| | Route de Presois 20 |
| | 1215 Geneva 15 |
| | Switzerland<br>Address |
| | Tel: +41 22 555 03 64 |
| | 101. 111 22 000 00 07 |

| | Email: gobeaun@mmv.org |
|---|---|
| Regulatory, Site Monitoring | Jolien Visser |
| and | Clinical Network Services (CNS) Pty Ltd |
| Data Management Functions | , , , |
| | ToowongQLD 4066, Australia |
| | Tel: +61 7 3719 6000 |
| | Email: Jolien.visse@clinical.net.au |
| Clinical Study Centre | Q-Pharm Pty Ltd |
| j | Level 5, 300C Herston Rd and |
| | Level 6, Block 8, Royal Brisbane and Women's Hospital |
| | Herston, QLD 4006, Australia |
| | Tel: +61 (0)7 3845 3636 |
| Clinical Laboratories | Clinical laboratory measurements |
| | Ms Marie-Claire Keogh |
| | Sullivan Nicolaides Pathology Central Laboratory (SNP) |
| | 24 Hurworth Street |
| | Bowen Hills, QLD 4006, Australia |
| | Tel: +61 (0)7 3377 8782 |
| | Email: marieclarie_keogh@snp.com.au |
| | Zmammano dano_koogn comprodimad |
| | Parasite quantification in blood samples |
| | Ms Jane Gaydon |
| | • |
| | Queensland Paediatric Infectious Diseases Laboratory (QP |
| | SASVRC, Level 8, Centre for Children's Health Research 62 Graham Street, |
| | South Brisbane, QLD 4101, Australia |
| | Tel: +61 (0)7 3069 7464 |
| | ` ' |
| | Email: j.gaydon@uq.edu.au |
| | Investigational drug quantification in blood samples |
| | Dr. Christoph Siethoff |
| | CEO |
| | Swiss BioQuant AG, |
| | Kägenstrasse 18 |
| | 4153 Reinach, Switzerland |
| | Email: Christoph.Siethoff@swissbioquant.com |
| | mail@swissbioquant.com |
| 0 : 45 : 450: | T +41 (0) 617 1698 12 |
| SeriousAE and AESI | Prime vigilance |
| reporting | Email:mmv@primevigilance.com |
| | Tel: +44 800 471 5694 |

# 2 INTRODUCTION: BACKGR OUND INFORMATION AND SCIENTIFIC RATIONALE

#### 2.1 BACKGROUND INFORMATION

Malaria is the second most prevalent infectious disease in the woorldthreaten shalf of the world's population. In accordance with the latest estimates by the World Health Organtison (WHO), there were an estimated 621 fillion new cases of malaria worldwide an 45,4000 deaths in 2016 [1]. The majority of these deaths were due to infection with falciparum. The WHO has declared malaria control a global development priority and has changed their recommendation from control programs to eradication programs.

Malaria drug resistance is a major hurdleatchievingmalaria eradication Resistance has been developed not only to conventional monotherapies such as chloroquine, amodiaquine and sulfadoxine/pyrimethaminebut also to the gold standard treatment for undicated P. falciparum malaria, artemisinin combination therapy (ACR) esistance to ACT's has been reported across the Greater Mek to region South East Asia [2, 3] and the inevitable spread of artemisinin resistance to Africa is of great concentremisinin resistance has been linked to mutations in the propeller domain of the falciparum Kelch 3 gene [4]. Artemisinin resistant isolates are not completely resistant at the misinin but instead have a slow parasite clearance phenotype compared to artemisision sitive isolates. This can lead to uced clearance of young ring-stage parasites, and therefore further maturation and sequestration of parasites leading to increased morbidity and mortality such a continual geometric future treatment options.

To achieve eradication of nalaria long-lasting, singledose treatments that completely clear malaria parasites from the body approvide a period of protection following the treatment are required These ideal types of medicines are defined to as singlencounteradical cure (SERC). The WHO and Medicines for Malaria Venture V(MV) have identified the key properties at a SERC must have. The seproperties are defined by Burroversal (2017) in the antimalarial target product profile (TPP)[5]. A key requirement of a target product is the inclusion two or more active molecules with different mechanisms of action the aim of including two or more active compounds is to achieve an increased barrier to resistance by using drugs with different mechanisms of action, forcing the parasite to develop medicipal ultaneous mutations in order to become resistant furthermore, a combination therapy, one of the two active compounds should have a rapid onset of action, killing most of the parasite IBarch active compounds should maintain plasma concentrationlevels above the minimal parasiticidal concentration (MIRC) approximately the same time and ensure complete elimination of all participates.

Artefenomel(OZ439), is a novel trioxolaneand afront-runner candidate for inclusion in a new antimalarial combination. It is a synthetic ozonide with potency comparable to artemisinin, with a rapid parasite clearance rate of approximately 3.6 Ph. ifalciparum Additionally, OZ439 has a substantiallylonger halflife than artemisinin (46 - 62 h as opposed to 3 h for artemisinin[6]). For these reasons, clinical studies in which artefenomel is combined with a companion drug with a differentmechanismof action are being planneour are currently in progress.

Piperaquine is ais 4-aminoquinoline and was used mainly in China from 1960's to the 1980's as an antimalarial monotherapy the 1980's, it became clear that parasite resistance developed to PQPmonotherapy PQP is characterise by slow absorption and a long elimination half-life (4–5 weeks) and is now widely used combination with dihydroartemisinin as a fixed dosed ACT. The successful paring of PQP with an artemisinin, together with biological half-life, means PQP is potentially a good drug partner for OZ439.

The safety, tolerability and PK profiles for OZ439 and PQP are well blished healthy subjects and in patients The antimalarial activity of the drugs individually sbeen demonstrated in IBSM studies in healthy subjects and in patients with uncompleted malaria. Phase Ib study of a single dose regimen of OZ439 800 mg in combination with 3 doses of PQP (640 mg, 960 mg, and 1440 mg) in adults and children with uncomplical educiparum malariahas been performed. Africa and Asia In this study, none of the dose arms of the study met the protocol health educive threshold of \$25\% based on the primary endpoint of polymerase chain reaction (ACDES) educate clinical and parasitological response (ACPR) outcome of Bolimythe per protocol analysis set. Therefore, an IBSM study assessing the antimalarial effect of OZ439 and PQP in a single dose combination could allow further understanding of the observed outcome of the OZ439 and PQP Phase IIb trial where treatment was also administered lingle dose combination.

Cumulatively, an estimated 1250 subjects have received OZ439 either alone or in combination with piperaquine phosphat(PQP), ferroquine (FQ) mefloquine, DSM265, or Cobicistat in clinical trials globally since the Development International Birth Datentil 29 March, 2018).

#### 2.2 RATIONALE

This study aims tevaluate the antimalarial activity of o-administered single doses of OZ439 and PQP in the IBSM model, and enable charactertiss of the exposure sponse relationship betweer OZ439 and PQP Pkind blood stage as exual parasitae Previous research has shown that the IBSM model is a good predictive model for real world antimalarial drug activity with single drug administratio [7]. However, it is yet to be determined if the model is an effective predictive tool when two or more drugs are administered in combination.

We hypothessie thatdata obtained a controlled diseaselike setting (Phase1 drugcombination IBSM model) carbe used to effectively redict the outcome of Phase 2studies in patients with uncomplicated malaria. To evaluate this hypothesis, we will assess if the trial can be used to predict what was observed in patients with uncomplicated malaria in the MMV\_OZ439\_13\_003 Phase 2b combination tr[8].

The doses chosen for use @nohort 1 are based on the APND relationships from the IBSM monotherapy studies and potential PD interaction effects of the combination based on the phase IIb study. Several doses will be tested in Cohort 1, which should achieve parasite reduction but not complete cure, such thatarasite regrowth can be observed, allowing an initial estimation of the PK/PD parameters of the 2 drugs when combined. The results of the first cohort will then be used to guide dose selection for Cohort 2 and simising the information on the PD interaction effect.

#### 2.3 POTENTIAL RISKS AND BENEFITS

#### 2.3.1 KNOWN POTENTIAL RISKS

Potential risks have been identified through review of previous clinical studies conducted to date using the IBSM modewith P. falciparum isolates as well as a review of the literature P. falciparum 3D7 has been sed to challeng \$12 healthy subjects 25 IBSM Phase thinical trials, 18 of which were successfully undertaken at QIMR Berghofe Poarm [9-34].

#### IBSM model risks

Risk management of blood borne infections

In this study,P. falciparum 3D7 inoculum will be used. This contains a very small amount of donor blood. However, the risk of infection from a possible blood borne virus from the blood transfused in this study tremely low for a number of reasons. Firstly, the donors were screened and tested negative of the presence of active blood borne infections. Secondly, white blood cells were removed from the donor blood by the Australian Red Cross Blood Service (Blood Service), which lowers the risk of transfusion transmitted infections. Thirdly, the volume of blood in the IBSM model for transmitting malaria is many thous of the smaller than in a transfused unit, thus reducing the risk of infection. As part of the safety monitoring, all subjects will have serum stored for testing of blood borne virus of the safety monitoring, all subjects who have received the P. falciparum 3D7 inoculum in IBSM studies.

Risk management of reaction to the blood sample

The risk of developingred blood cell (RBC) alloantibodies in this study is considered extremely low since the donor blood used to produce ithous ulant was blood group O R(D) Negative.

People with this blood group are generally considered "universal donors", as recipients of their blood have minimal risk of developing RBC alloantibodies when given much larger volumes of blood than is used in the IBSM model. However, it is possible that subjects could suffer a transfusion reaction after they receive the inocular develop alloantibodies to the donor RBCs that may make blood transfusion more difficult in the future. To date, one subject has developed an antibody response to a minor Rh antigen (antitibody) following inoculation with falciparum 3D7 [35]. However, there was no laboratory evidence to indicate that the specific R phenotype of the donor RBCs in the inoculum provoked production of this all antibody. Subjects will be monitored for signs and symptoms in the period immediately after administration of the inoculum to further assess the risk of the inoculura insing a transfusion reaction. Subjects will also be tested for RBC alloantibodies at screening and at the end of the study as part of their safety monitoring Section 7.2.1)

Women of childbearing potential (WOCBP) have a small additional riskten/eloping RBC alloantibodies that could cause problems during preacy. WOCBP have participated in several IBSM trials with P. falciparum isolate 3D7 with no known issues to date. Specific strict contraception requirements will be requested for this patiput during the study/Section 5.1.) Including WOCBP in the trial enhances the generalisability of the study results.

#### Risk management of malaria infection

The number of viable blood stageparasites used to infect the subjects in this stud(y-2,800) is substantially lower than the parasitaemia reached after the bite of a single malaria-infected mosquito, where approximately 30,000 parasites are released into the blood when they break out of a single infected liver cell [36]. In this study, parasite growth malaria symptoms will be closely monitored in subjects following administration of the challenge agreenth reshold for commencement of antimalarial drug reatment defined for this study (2) (ay 8) has been selected since it is prior to the timepoint at which advanced clinical symptoms of malaria are likely to occur, as observed in the previous 25 clinical trials performed with the 3D7 challenge agent.

#### Risk management of liver functionabnormalities

Transient, asymptomatic liver function test (LFath)normalities including rare cases calanine aminotransferascent aminotransferascelevations >100ld theupper limit of norma(xULN) have been reported in several subjects in IBSM stutes and included in several subjects in this stude and included included in several subjects in this stude and included in several subjects in this stude and included in several subjects in this stude and included in several subjects in this stude and included included in several subjects in this stude and subjects in this stude and su

safety monitoring to assess for asymptomatic LFT abnormalities. Subjects are required to intake of possibly hepatotoxic substances as alcoholand paracetamoduring the course of the study (see Section 5.2 & 7.6). Drugs of abuse are not permitted under any circumstance.

#### Risk management of cardiacAEs

To our knowledge, & ardiacSAEs have been reported in healthy subjects in the Netherlands participating in malaria challenge studies using sporozoites i.e. direct feeds by infected mosquitoes rather than IBSM infectionRefer to the P. falciparum3D7 Investigators Brochures for further details[35]. No cardiac SAEs caused by the inoculum have beported in IBSM studies. As a precaution, people at significant risk of cardiovascular disease will be excluded from participating in IBSM studies, and regular safety monitoring including physical examination and electrocardiogramE(CG) recordings will the place for all subjects.

# Investigational Medical Product (IMP) risks

#### OZ439 risks

To date, OZ439 administered either as a monotherapy or in combination with a partner anti malarial, has been generally well tolerated in malaria patients in the althy sujects. In a monotherapy Phase IIa study of OZ439 doses of 200, 400, 800 and 1200 mg in malaria patients, increased blood creatine phosphokinase was the most frequently repetited; a dose relationship was not seen for this Astend no clinically relevant muscular AE were reported. Gastrointestinal (GI) AEs, including vomiting, abdominal pain, diamaheand nervous system disorders, including dizziness and headache, were reported more frequently with 1200 mg OZ439 compared to the other dose cohorts. Note that the compared to the other dose cohorts. Note that the compared to the other dose cohorts.

One case of vasvagal syncope considered related to therapy was reported in association with sinus arrest and orthostatic hypotension. Two SAEs of atrial fibrillation were reported in healthy volunteers. One case occurred at day 35 post dose and waiseidless not related to the study drug. The second case was moderate atrial fibrillation, considered sibly related to the study drug in a subject who had received OZ439 and FQ. The event occurred in context of symptomatic orthostatic hypotension and solved spontaneously without medical treatment.

In a Phase IIb study, where OZ439 was evaluated in combination with PQP, in patients with uncomplicated P. falciparummalaria, malaria and electrocardiogram (ECG) QTc prolongation were the most frequent protect AEs. Malaria was reported with a higher incidence in the OZ439 800 mg:PQP 960 mg and in the OZ439 800 mg:PQP 640 mg treatment arms than in the OZ439 800 mg:PQP 1440 ng treatment arm. The ECG QTc prolongation was reported with a higher incidence in the OZ439800 mg:PQP 1440 mg and the OZ439 800 mg:PQP 960 mg treatment arms than in the OZ439 800 mg:PQP 640 mg treatment arm. Concentral at the OZ439 800 mg:PQP 640 mg treatment arm.

has been widely documented with PQP. Dianthend vomiting were the most frequently netpd AEs of the GI system in patients treated with both OZ439 and PQP. None of these AEs were SAEs.

The AE profile for OZ439 in healthy subjects was similar to the AE profile in malaria patients. Gastrointestinal AEs, including nausea, vomiting, and lower, were the most frequently reported AEs in healthy subjects treated with OZ439 alone or OZ439 in combination with either PQP, MQ, or FQ. A tendency for a dosesponse relationship was seen for GI ever the every series of the every se

Eight subjects treated with OZ439, including 6 malaria patients and 2 healthy volunteers, have had SAEs, including P. vivax relapse, pyelonephritis, increased alanine aminotransferase (ALT), increased aspartate aminotransferase (AST), decreased neutrophit, anemia, febrile convulsion and decreased hemoglobin in malaria patients; and atrial fibrillation and a gunshot wound in healthy subjects. Fir AEsreported malaria patient (increased ALT, increased AST, decreased neutrophil count, anemia and decreased hemoglobin) were assessed as related to study drug by the investigator

An AE of vomiting led to study drug discontinuation in 1 malaria patient treated with OZ439. Ten healthy subjects treated with OZ439 discontinued a Phase Ia study due to an AE. Vomiting (5 subjects) was the most frequently reported AE leading to study discontinuation in the 10 healthy subjects. Except for a few cases observed with  $\alpha$ -tocopherol polyethylenglycol 1000 succinate (TPGS) formulation, vomiting is not reported in healthy subjects at doses < 800 mg OZ439.

No Hy's law cases have been observed. However, mild to severe and reversible increases in ALT and AST were seen in OZ43@cated malaria paties, these increases did not appear to be-dose dependent. Decreases in hemoglobin, neutrophils, and platelets were also seen itreated malaria patients; however, these decreases were consistent with those observed in acute malaria. Close monitoring bliver function is required in the clinical studies.

In the clinic, a significant effect on placeborrected change from baseline QTcF was not demonstrated for OZ439. In healthy subjects the effect of OZ439ng0@lone on QTc was minimal, with a maximummean QTcF increase from baseline and placebo ofm8.5 (StudyMMV\_OZ439\_12\_002). In Study MMV\_OZ439\_12\_003, 1 healthy subject with an undisclosed history of mitral and tricuspid regurgitation was discontinued from the study due to asymptomatic supraventrilar/junctional tachycardia after dosing with 120 mg OZ439. QTc prolongations (both QTcB and QTcF) were seen when OZ439 was administered in combination with PQP to malaria patients and healthy subjects. Most of the prolongations were in the range of >30 ms but <60ms; however, prolongations >60 ms were observed in malaria patients, with QTcF values that exceeded 500 ms in 2 patients (1 hypokalemic patient). Reversible right bundle branch block (3 patients), reversible first degree atrioventricular blogba(fent), and a mild reversible

sinus bradycardia (1 patient) were also observed in malaria patients treated with OZ439. Close monitoring of cardiac function is required in the clinical studies.

In healthy subjects treated with OZ439 alone or OZ439 inbovention with PQP, gastrointestinal (GI) symptoms which include nausea, vomiting, and diarrhea, are the most commonly reported AEs and these AEs haveen reported to be generally mild in intens 22/2439 was clinically well tolerated intwo previous IBSMstudies(QP12C10 and QP14C12) here the highest dose tested was 500 mg. In a Phase IBBSM study QP12C10 in healthy subjects infected Withalciparum most of the AEs reported were assessed as probably related to the inoculum (i. e., malaria). There were no events considered probably related to OZ439ndrtherPhase IBBSM study QP14C12. healthy subjects infected with falciparum received OZ439in combination with another investigational antimalaria DSM265 No new clinically relevant safety signals were observed. OZ439 may be contraindicated in persons with known hypersensitivity to artembaissed compounds or to any components of the product formulation. Carcinogenicity studiesohave been performed whit OZ439.OZ439 has shown in vivo embrifetal toxicity in the rat. Therefore, OZ439 shouldnot be administered to pregnamtbreastfeedingwomen. However, OZ439anbe administered to women of child bearing potential (WOCBP) thichuse of strictdouble method of contraception well controlled clinical trials and under medical supervisities althy male and female subjects participating in studies of OZ439 must agree to use a double method of contraception for a duration defined in section (5) clusion criteria) of this protocol.

No deaths have been reported by of the clinical studies.

Additional information on nominical and clinical studies conducted with OZ439 is provided in the IB[38].

#### Piperaguine phosphate(PQP) risks

PQPas a combination antimalarial withhydroartemisiniris well tolerated both adults and children, with the main AEs reported bing GI disturbances such as diarrh [69, 40]. Studies with dihydroartemisinin PQP demonstrated corrected QT (QTc) interval prolongation during treatment [41, 42]. Very few individual patients ave been observed to have prolongation that could be regarded as clinically sigcant (>60 msec); of note, the QTc prolongation induced by PQP hasnot been reported to be associated with clinically relevant cardiovascular evolutions, would suggest lack of pro-arrhythmic effect. Therefore, although statistically significant, the QTc prolongation observed following Ptherapy is unlikely to be of clinical concern. European regulatory authorities have advised that Eurart esitalihydroartemisinin PQP) not be administered with food to redude Ppeak concentrations, and caution the ibraior and post electrocardiographic monitoring be undertaken, and avoidance of concomitant recent exposure to drugs at risk of QTc prolongation and will have ECGs recorded before and after treatment.

PQPhas beenclinically well tolerated previous IBSM studies using this dr[64]. In these studies, PQP treatment demonstrated robust safety profile in doses up to 960 mg when used for the treatment of uncomplicated falciparummalaria infection.

Details on the safety and efficacy of PQP as part of the combination product Eurarteainbe found in the European Medicines Agen&M(A) European Public Assessment Report.

#### Rescue Medication risks

Riame<sup>®</sup>, Primacir<sup>™</sup> and Artesunateisks are detailed in their respective approved manufacturer's prescribing information (Appendix 1). Primacin may cause severe haemolytic anaemia in subjects with glucose-phosphate dehydrogenase (G6PD) deficiescybjects will be tested for G6PD deficiency at screening to ensure the safety of Primacin<sup>™</sup>. The G6PD status will determine how the subject is treatevith Primacin<sup>™</sup>.

#### General risk management

The risk tosubjects this study will also be minimised as follows:

- Adherence to the inclusion/exclusion criteria to ensure that only subjects whotære any perceived risk are enrolled in the study
- Close clinical and laboratory monitoring to ensure the safety and by and
- Subjects will be prescribed curative therapy for malaRiamnet® with the addition of Primacin<sup>TM</sup> if required) for final parasiteclearance during or at the end of thedstu
- The total volume of blood drawn from each subject enrolled into the study (including optional exploratory research sampling) will not exceed a standard unit of blood (approximately 450 mL) over any 30ay period.
- In the rare event that a subject requi hospitalisation at the request of the Principal Investigator his representative, this will be done the Infectious Diseases Unit, Royal Brisbane and Women's Hospital. Emergency procedures are in place at the Q-Pharm clinics for dealing with any unforeseen clinical emergencies which may arise.

With these safety provisions, the overall risk to the subjects in the study is considered to be minimal and acceptable, and the potential of future improved treatment for malaria is considered to outweigh these potential risks.

#### 2.3.2 KNOWN POTENTIAL BENEFITS

There is no expected clinical benefit for the healthy subjects that will participate in this study. Overall, on the basis of the available redimical and clinical data, and prior knowledge, the risk benefit profile of OZ439 and QPare judged acceptable for the proposed clinical study.

# 3 OBJECTIVES AND PURPOSE

### Primary:

- a) To characterize the PK/PD relations this tween OZ439 and PQP lasma concentrations and blood stage as exupatrasita emian healthy subjects following. falciparum IBSM infection.
- b) To evaluate the safety and tolerability of OZ439 and PQP whendronistered as single doses in healthsubjects following falciparum IBSM infection

## Secondary:

- a) To describe the PK of OZ439 and PQP wheradministered as single doses in healthy subjects under fasted conditions.
- b) To characterize the PD effect of-administered single doses of OZ439 and PQP on clearance oP. falciparumasexual blood stage parasites from the blood of healthy subjects in the IBSM model.

## **Exploratory**:

The exploratory study objectives are:

- a. To characterise specific cell subsets and immune signatures associated with control of parasite burden and pathogenicity following first exposure to P. falciparum, to identify specific cells, immunomodulatory molecules and immunehways to target for therapeutic intervention.
- b. To investigate the role of RBC complement regulatory proteins and anti phosphatidylserine antibodies in malarial anaemia.
- c. To investigate the association between serum complement activation, complement activating antibodies, and RBC complement regulatory protein expression.

#### 4 STUDY DESIGN AND ENDPOINTS

#### 4.1 DESCRIPTION OF THE \$UDY DESIGN

This is a singlecentre, open label, adaptive study using the P. falciparum IBSM inoculum as a model to character is the PD activity of combined administration of OZ439 and PQP

The study will be conducted in a maximum of three cohorts (up to 8 subjects per cohort) using up to 4 different doses of OZ439 and PQP in each cohos ubjects will be malariana ve healthy males of females aged between 185 years old, who meet all of the inclusion criteria anothe of the exclusion criteria Additionally, the study includes ptional, exploratory components, which require separate informed consent for subjects agreeing to participate in these.

The first cohort will comprise groups of subjects each subjects will be administered single oral doses of OZ439 and PQP in combination. The dose 4892 and PQP will be different for each group in Cohort 1, and subjects will be randomised into one of the dose groups listed in Table 1.

Table 1 OZ439 and PQP Cohort 1 Dose

| Drug | | Dose group | | |
|-----------|-----|------------|-----|-----|
| | 1A | 1B | 1C | 1D |
| OZ439(mg) | 200 | 200 | 400 | 400 |
| PQP(mg) | 480 | 640 | 480 | 640 |

The data captured from this first cohort will be used to determine the relationship belowed and PQP concentrations and parasitaemia levelsed onsafetyandtolerability data up to Day 42±2 and PK/PDanalysis outcomes (based on PD data up to 422±2 and PK data up to as 35±2), of the drugs given in combination dos(s) for the subsequent cohort will be determined

After review of the PK/PD and safety data from Cohort 1 by SDRT it was determined that, the second cohort will be composed of 2 dose groups of 4 subjects Seatophects will be randomised into one of 2 dose groups and administered single oral doses of OZ439 and PQP in combination The combined dose 60Z439 and PQP will be different for each group in this cohort as shown in Table 2.

Table 2 OZ439 and PQP Cohort2 Dose

| Drug | Dose | se group |
|-----------|------|----------|
| | 2A | 2B |
| OZ439(mg) | 800 | 200 |
| PQP (mg) | 960 | 320 |

A similar analysis will be done at the end of cohort 2 combining control 2 data to decide the dose(s) to be tested in cohort 3. This will be decide they funding sponso and the Principal Investigator following SDRT and scientific evaluation

The doses used in all Cohorts will not exceed 800 mg for OZ439 and 1440 mg for PQP as determined in previous safety, pilot efficacy and phase 2 stubbles subject will be inoculated on Day 0 with approximately 2,800 vilatoparasites of P. falciparum infected human erythrocytes administered intravenously Subjects will be monitored daily via phone call text messagen Days 1 to 3 positoculation to solicit any AEs.

Then, subjects will come to the clinical unit ordaily basisfrom Day 4 until the presence of asexual parasites is established PCR targeting the 18S rRNA gene (referred to as malaria 18S qPCR). Once qPCR becomespositive and until OZ439 and PQP administration subjects will attend the clinical unit fotwice-daily visits, separated by approximately 12 hours, for clinical evaluation and blood sampling.

Subjects will be admitted to the clinical unit fixingle dose administration 67Z439 and PQP 8 days after malaria inoculation earlier if a subjecthas amalaria clinical score >60r at Investigators discretion An intravenous cannula will be placed and preliminary blood samples collected. The participants will then baselministered the IMP in a fasting statemmediately Subjects in the first cohomnay all be dosed on the same days eithese exposures have been documented previous studies and shown to be well tolerated.

Once single dose candministration of OZ439 and PQP occurrebjectswill be followed up as inpatients for at least 72 hours thonitor for safety and tolerability of the treatment and to ensure adequate clinical and parasitological tesponse Blood samples will be collected poses and following OZ439 and PQP reatment to measure plasma concentration SZ439 and PQP. Wherever possible, PK sampling will coincide with postose blood collection for monitoring of parasitaemia.

After 72 hours, if clinically well, subjects will be discharged from the clinical unit and will be followed up regularly for safety assessments, PK sampdingical evaluation and malaria qPCR blood sampling untilDay 42±2. All subjects will receive a standard course of therapy with

Riamet® (artemethelumefantrine) on Day 422 or earlier in the event of failure of clearance of parasitaemia defined as failure to clear parasitaemia by at leastott 72 hours postMP administration Riamet will also be administered in the eventrecrudescence of parasitaemia (definedas ≥5 000 blood stage parasites/mL and a 2-fold increase within 48 hours, or a malaria clinical score >6 or at Investigatos discretion. If indicated by the presence of gametocytes at the time of treatment with Riamet®, Primacin<sup>TM</sup> 45 mg will also be administered as a single oral dose.

Subjects participating may optionally consent to be included in the exploratory components of the studywhich require additional blood samples to be collected at specifieebtoinness throughout the study. These timeoints coincide with those already scheduled as part of the main study assessments. If any of the main study timoents change the exploratory study timoents will change to match Details of the exploratory components and analyses are provident of the study timoents.

A review by the SPRT of data from each cohort will be conducted prior to dosing the subsequent cohort. Safety and tolerability data up toDay 42±2 and PK/PDanalysis outcomes (based on PD data up to Day 42±2 and PK data up toDay 35±2), from all subjects who received eatment with OZ439 and PQP will be required for the review similar analysis will be done at the end of cohort 2 combining cohort 1 and 2 data to decide the decided by the funding sponsor and Primercipal Investigator following review of the data by the SDRT and scientific evaluation.

The doses used in all cohorts will not exceed the maximum acceptable doses predefined for this study (800 mg for OZ439 and 1440 mg for PQP) as determined in previous safety(fipitoty and phase 2 studies.

#### 4.2 STUDY ENDPOINTS

#### 4.2.1 PRIMARY ENDPOINT

- The PK/PD relationship between OZ439 and PQP plasma concentrations and blood stage asexual parasitaemia will be determined by:
  - Effect of OZ439 on Fax and EG<sub>0</sub> of PQP
- The safety and tolerability of a single combined dose of OZ439 and PQP will be evaluated by the incidence, severity and relationship of observed and expelfted AEs up to trial Day 42±2 after the co-administration of single doses of OZ439 and PQP to subjects inoculated with IBSM.

#### 4.2.2 SECONDARY ENDPOINTS

- Estimation of OZ439 and PQP PK parameters trial Day 422 after coadministration of single doses using nonempartmental nethods: AUG-168h, AUClast, AUCO-inf, Cmax, tmax, t<sub>1/2</sub>, t<sub>lag</sub>, C<sub>168h</sub>, CL/F, Vz/F and λ<sub>inf</sub>.
- The effect of coadministered single oral doses of OZ439 and PQP on clearance of P. falciparumblood stage parasitesom the blood of inoculated subjects as measured by qPCRup to trial Day 422 after coadministration of OZ439 and PQP. Parasite clearance will be assessed by the following parameters:
  - Parasite clearance hailfe (Pt ½).
  - Parasie reduction ratio (PRR)
  - o Percentage of subjects with recrudescence of parasitater fine das≥5 000 blood stage parasites/mL and afo2d increase within 48 hours, or-occurrence of malaria symptoms with a malaria clinical score.>6)

#### 4.2.3 EXPLORATORY ENDPOINTS

- Identification of immune checkpoint molecules.
- The level of expression of complement regulatory proteins (CD35, CD55 and CD59) and phosphatidylserine on RBC.
- The levelof complement activating antibodies and aptrosphatidylserinantibodies.

# 5 STUDY ENROLLMENT AND WITHDRAWAL

#### 5.1 SUBJECT INCLUSION CRITERIA

Subjects eligible for inclusion in this study must fulfil of the following criteria:

#### Demography

- 1. Adult (male and emale) subjects between 18 and 55 years of age inclusive, who do not live alone (from inoculation day until at least the end of Riemet® treatment) and will be contactable and available for the duration of the trial and contactable up to 2 weeks following the End of Study visit (approximate% 5 weeks).
- 2. Body weight minimum 50 kg, body mass index between 18 and 32, kig/thusive.

#### Health status

- 3. Certified as healthy by a comprehensive clinical asses (detailed medical history, complete physical xamination and special investigations
- 4. Vital signs after 5 minutes resting in supine position:
  - 90 mmHg  $\leq$  systolic blood pressure (SBP)  $\leq$  140 mmHg,
  - 40 mmHg  $\leq$  diastolic blood pressure (DBP)  $\leq$  90 mmHg,
  - 40 bpm  $\leq$  heart rate (HR)  $\leq$  100 bpm.
- 5. Must have QTcF ≤450 ms, QTcB ≤450 ms for male subjects, QTcF ≤470 ms, QTcB ≤470 ms for female subjects and PR interval ≤210 msat screening and at prenoculation or day.
- 6. Heterosexualwomen of childbearing potential should be surgically sterile or using an insertable, injectable, transdermal or combination oral contraceptive approved by the TGA combined with a barrier contraceptive for the duration of the study, and have negative results on a urine pregnancy test done befoire culation Abstinent, heterosexual reale subjects must agree to start a double method if they start a sexual relationship during the study. Adequate contraception does not apply to subjects of childbearing potential with same sex partners (abstinence from penileginal intercourse), when it is their preferred and usual lifestyle. Female subjects with same sex partners must not be plain viritgo fertilisation within the required contraception period.

Women of norchildbearing potential who will not require contraception during the study are defined as: postnenopausal (spontaneous amenorrhoea for  $\geq 12$  months, or spontaneous

amenorrhoea for -62 months and follicle timulating hormone (FSH)  $\geq$  40 IU/mL; either should be together with the absence of oral contraceptive use for > 12 months).

Male subjects participating must agree to use a debutableer method of contraception including condom plus diaphragm or condom plus intrauterine device or condomstables oral/transdermal/injectable hormonal contraceptive by the female pairtonnerthe time of informed consenthrough to 90 daysafter the last dose © Z439 and PQPAbstinent male subjects must agree to start a doubtakerier method if they begin seems relationships during the study and up to 90 days after the last dose of study drug.

Male subjects with female partners that are surgically sterilemale subjects who have undergone sterilisation and have had testing to confirm the success efitisation may also be included.

# Regulations

- 7. Having given written informed consent prior to undertaking any stellaged procedure.
- 8. Must be willing and able to communicate and participate in the whole study.

#### 5.2 SUBJECT EXCLUSION CRITERIA

Subjects fulfilling any of the following criteria will not be eligible for inclusion in this study:

Medical history and clinical status

- Haematology, clinical chemistry, coagulation or urinalysis results at screening or on admission prior tonoculation or IMP administration that are outside of Sponapproved clinically acceptable laboratory ranges documenited the laboratory manual are considered clinically relevant.
- 2. Any history of malaria or participation in a previous malaria challenge study.
- 3. Must not have travelled to or lived (>2 weeks) in a malæriædemic region during the past 12 months or planned travel to a malæriædemic region during the course of the study (for endemic regions selettps://map.ox.ac.uk/countpyrofiles/#!/). Bali is not considered a malariaendemic region.
- 4. Participation in any investigational product study within the 12 weeks preceding administration
- 5. Has evidence of increased cardiovasculls at serisk (defined as >10%y far risk for those greater than 35 years of agas determined by the Australian Absolute Cardiovascular Disease Risk Calculato http://www.cvdcheck.org.a))/. Risk factors include sex, age,
- systolic blood pressure (mm/Hg), smoking status, total and HDlesslevol (mmol/L), and reported diabetes status.
- 6. Symptomatic postural hypotension at screeningwoconsecutive readingis respective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 2-3 minutes when changing from supine to standing position.
- 7. History of splenectomy.
- 8. History or presencefoliagnosed (by an allergist/immunologist) or treated (by a physician) food or known drug allergies (including but not limited to allergy to any of the antimalarial rescue medications to be used in the study), or history of anaphylaxis or other serogice alle reactions. Note. Subjects with seasonal allergies/hay fever, house dust mite or allergy to animals that are untreated and asymptomatic at the time of dosing can be enrolled in the study
- 9. History of convulsion (including intravenous drug or vacaimeuced episodes) Note. A medical history of a single febrile convulsion during childhood is not an exclusion criterion.
- 10. Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immunateficiencies), insum-dependent and nansulin dependent diabetes (excluding glucose intolerance if exclusion criterion 4 is met), progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, porphyria, ripassis, rheumatoid arthritisasthma, epilepsy, or obsessive compulsive disorder.
- 11. History of malignancy of any organ system (other than localised basal cell carcinoma of the skin orin situ cervical cancer), treated or untreated, within 5 years of screening ardless of whether there is evidence of local recurrence or metastases.
- 12. Subjects with history of schizophrenia, phoilar disease, or other severe (disabling) chronic psychiatric diagnosis including depression or receiving psychiatric drugs or whomehas hospitalised within the past 5 years prior to enrolment for psychiatric illness, history of suicide attempt, or confinement for danger to self or others.
- 13. History of serious psychiatric condition that may affect participation in the study or preclude compliance with the protocol, including but not limited to past or present psychoses, disorders requiring lithium, a history of attempted or planned suicide, more than one previous episode of major depression, any previous single episode of major depressio lasting for or requiring treatment for more than 6 months, or any episode of major depression during the 5 years preceding screening.

The Beck Depression Inventory (Appendit) will be used as an objective tool for the assessment of depression at sciregen addition to the conditions listed above, subjects with a score of 20 or more on the Beck Depression Inventory and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation) will not be eligible for participation. These subjects will be referred to a general practitioner or medical specialist as appropriate. Subjects with a Beck score of 17 to 19 may be enrolled at the discretion of the secution of the subject or to the execution of the study and interpretation of the data gathered.

- 14. History of recurrent headache (e.g. tenstigme, cluster or migraine) writa frequency of  $\geq 2$  episodesper month on averagend/orsevere enough to require medical therapy.
- 15. Presence of acute infectious disease or fever (e.g. sublingual temperature ≥38.5°C) within the 5 days prior to inoculation with malaria parasites.
- Evidence of acute illness within the 4 weeks prior to screening that vtbstigatordeems may compromise subject safety.
- 17. Significant intercurrent disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmudisease by history, physical examination, and/or laboratory studies including urinalysis.
- 18. Subject has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion (e.g. gastrectomy, diarrhoea)
- 19. Blood donation of any volume within 1 month before inclusion, or participation in any research study involving blood sampling (more than 450 mL/unit of blood), or blood donation to Australian Red Cross Blood Service (Blood Service) or other blood brands du the 8 weeks prior to the treatment drug dose in the study.
- 20. Subject unwilling to defer blood donations to the Blood Service for at least 6 months.
- 21. Medical requirement for intravenous immunoglobulin or blood transfusions.
- 22. Subject who has ever receive black transfusion.
- 23. History or presence of alcohol abuse (alcohol consumption more than until 4 standard drinks per day) or drug habituation, or any prior intravenous usage of an illicit substance.
- 24. Tobacco use of more than 5 cigarettes or equiv**plend**ay, and unable to stop smoking for the duration of the clinical unit confinement.
- 25. Female subject who is breastfeeding.

# Interfering substances

- 26. Any vaccination within the last 28 days.
- 27. Any corticosteroids, antinflammatory drugs, immunomodulators ontiacoagulants. Any subject currently receiving or having previously received immunosuppressive therapy (including systemic steroids, adrenocorticotrophic hormone or inhaled steroids) at a dose or duration associated with hypothalanpiituitary-adrenal axissuppression (e.g. 1 mg/kg/day prednisone, chronic use of inhaled high potency corticosteroids such as budesonide 800 μg/day or fluticasone 750 μg, or equivalent).
- 28. Any recent (<6 weeks) or current systemic therapy with an antibiotic or drug with potential antimalarial activity (e.g. chloroquine, piperaquine phosphate, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, doxycycline etc.).
- 29. Ingestion of any poppy seeds within the 24 hours prior to the screening blood test (subject will be advised by phone not to consume any poppy seeds in this time period).
- 30. Excessive consumption of beverages or food containing xanthine bases including Red Bull, chocolate, coffee etc. (more than 400 mg caffeine per day, equivalent to more than 400 mg caffeine per day).
- 31. Unwillingness to abstain from consumption of grapefruit or Seville oranges from inoculation day until end of the study
- 32. Unwillingness to abstain from consumption of quinine containing foods/beverages such as tonic water and lemon bitter, from inoculation day until entainer treatment.
- 33. Use of prescription drugs or nonescription drugs or herbal supplements (such as St John's Wort), within 14 days or 5 halfves (whichever is longer) prior to the malaria inhaction. As an exception, ibuprofen (preferred) may be du at doses of up to 1.2 g/day paracetamol at doses of up to to to the romprescription medications or dietary supplements, not believed the test subject safety or the overall results of the study, may be permitted on to the study approval by the Sponsor in consultation with the estigator Subjects are requested to refrain from taking nonapproved concomitant medication recruitment until the conclusion of the study.

#### General conditions

34. Any subject who, in the judgment of the vestigator is likely to be nor compliant during the study, or is unable to cooperate because of a language problem or poor mental development.

- 35. Any subject in the exclusion period of a previous study according to applicable regulations.
- 36. Any subject who is the Principalnestigator any subinvestigator research assistant, pharmacist, study coordinator, or other staff thereof,cdirenvolved in conducting the study.
- 37. Any subject without a good peripheral venous access.

# Biological status

- 38. Positive result on any of the following tests: hepatitis B surface antigen (HBs Ag), anti-hepatitis B core antibodies (art Bc Ab), anti-hepatitis C virus (ant HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (art 1 and anti-HIV2 Ab).
- 39. Positive urine drug test. Any drug listed in Section 7.2.1 in the urine drug screen unless there is an explanation acceptable to **the**estigator(e.g., the subject has stated in advance that they consumed a prescription or owner product which contained the detected drug) and/or the subject has a negative urine drug screen on retest by the pathology laboratory. Any subject testing pitive for acetaminophen (paracetamol) at screening may still be eligible for study participation, at the vestigators discretion.
- 40. Positive alcohol breath test.

### Specific to the study

### 41. Cardiac/QT risk:

- Family history of sudden death or of congenital pmglation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
- History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.
- Electrolyte disturbances, ptianularly hypokalaemia, hypocalcaemia, or hypomagnesaemia.
- ECG abnormalities in the standard-le2d ECG (at screening at preinoculation on inoculation da) which in the opinion of thenvestigatoris clinically relevant or will interfere with the ECG nalyses.
- 42. Known hypersensitivity to artesunate or any of its excipients, artemether or other artemisinin derivatives, piperaquine phosphate, proguanil/atovaquone, primaquine, -or 4 aminoquinolines.

Healthy subjects who do notalfil all the inclusion criteria, and/or fulfil any of the exclusion criteria should not be enrolled into the study without exception. In case of doubtyelseigator is to confer with the medical monitor for agreementativers for inclusion of volunteers that are not meeting all edibility criteria will not be granted

Subjects who are excluded from participation on study days for any of the abovereasons may be eligible to participate on a postponed schedule, if the Investigator considers this appropriate.

#### 5.3 CONTRACEPTION

Male and female subjects who are sexually active must use, with their partner, 2 approved methods of highly effective contraception from the time of informed consent until 90 altays the last dose of OZ439 and PQP.

Two or more of the following methods arecaptable and must include at least 1 barrier method:

- Surgical sterilisation (vasecton(male), tubal ligation (female)
- Placement of an intrauterine device or intrauterine system
- Hormonal contraception (implantable, patch, oral, injectable)
- Barrier methods (this must be a condom or their partner's use of an occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository)

Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, they, with their partner, must comply with the contraceptive requirements detailed above.

Adequate contraception does not apply to subjects of childbearing potential with example theres (abstinence from penile aginal intercourse), when this is their preferred and usual lifestyle. Female subjects with same sex partners must not be plaim in for fertilisation within the required contraception period.

Women of norchildbearing potential who will not require contraception during the study are defined as: postnenopausal (spontaneous amenorrhoea for  $\geq 12$  months, or spontaneous amenorrhoea for 6-12 months and folliclestimulating hormone (FSH)  $\geq 40$  IU/mL; either should be together with the absence of oral contraceptive use for > 12 months) or permanently sterilised (e.g. hysterectomy, bilateral salpingectomy).

Adequate contraceptions also not required formale subjects with female partners that are permanently sterilised male subjects who have undergone sterilisation and have had testing to confirm the success of the sterilisation.

#### 5.4 STRATEGIES FOR RECRUMENT AND RETENTION

Up to 24 subjects are planned to be enrolled in the study. It is estimated that approxi76 ately subjects may need to be screened to complete enrolled in the study. It is estimated that approxi76 ately subjects may need to be screened to complete enrolled in the study. It is estimated that approxi76 ately subjects may need to be screened to complete enrolled in the study. It is estimated that approxi76 ately subjects may need to be screened to complete enrolled in the study. It is estimated that approxi76 ately subjects may need to be screened to complete enrolled in the study. It is estimated that approxi76 ately subjects may need to be screened to complete enrolled in the study.

Subjects will be recruited from the QIMR Berghofer Human Research Ethics Committe® (QIM Berghofer HREC) approved database of healthy subjects maintaine® by not on by a general or study specific advertisement via print, radio or poster media to students of Queensland universities or to the general community, as approved by the QIMRh® mergHREC. No restrictions will apply for ethnic or racial categories; the expected population may include all Australian racial categories.

Subjects who complete the study up to Asy2/EOS will be paid\$3,865compensation for their participation. Subjects who withdraw or are withdrawn from the study will be compensated on a fractional basis for their involvement unless they are withdrawn as a consequence of their misconduct. Reserve subjects who do not participate in the study will b\$150dompenation (per inoculation day) for the inconvenience associated with their attendance for screening and for their attendance on the inoculation day, in case they are required to participateers who fail screening due to an underlying medical conditions viously unknown to them will be reimbursed \$75 for their time, and provide with the appropriate referrals for guidance and counselling fortheir condition.

#### 5.5 SUBJECT WITHDRAWAL OR TERMINATION

### 5.5.1 REASONS FOR WITHDRAWAL OR TERMINATION

Subjects are free to withdraw from the study at any time. A subject may be considered withdrawn if he/she states an intention to withdraw, fails to return for scheduled protocol visits for any reason, or becomes lost to followp. Subjects may also be withawn by thenvestigator Possible reasons for withdrawal by thenvestigatorinclude the occurrence of SAE, failure by the subject to comply with the requirements of the protocol, or for any other reason at the discretion.

# 5.5.2 HANDLING OF SUBJECT WITHDRAWALS OR TERMINATION

If a subject is withdrawn from the study, the funding Sponsor will be informed immediately. If there is a medical reason for withdrawal, the subject will remain under the supervision of the Principal Investigatountil satisfactory health has returned.

The Investigatorwill make every effort to determine the primary reason for a subject's withdrawal from the study and record this information in the electronic case report form (eCRF). For subjects who are lost to follow-up, the Investigatorwill demonstrate due diligence by documenting all steps taken to contact the subject (e.g. dates of phone calls, registered letter, home visit, etc.) in the source documents. If earlier withdrawal from further study procedures of the Issubject will be asked to complete the antimalarial rescue treatment. The subjects will also be asked to complete the early termination evaluation as described in Section 7.3.5.

If the subject is withdrawn from the study procedures or followfor any reason, with the subject's permission, medical care will be provided for any SAEs that occurred during participation in the study until the symptoms of any SAEs are resolved and the subject's condition becomes stable. Followp for AEs is described in Steon 8.3.

If a subject is withdrawn due to a study dragated AE or due to termination of the study, the early-termination subject will not be replaced. If a subject does not complete the study for reasons other than safety, the early termination subject may become after mutual agreement between the funding Sponsor and three-vestigator The decision regarding the replacement of subjects will be documented.

### 5.6 PREMATURE TERMINATION OR SUSPENSION OF BUDY

The Sponsor, Principalnvestigator QIMR Berghofer HREC and Regulatory Authorities independently reserve the right to discontinue the study at any time for safety or other reasons. This will be done in consultation with the Sponsor where practical. In the event of premature trial termination or suspension, the bovementioned parties will be notified in writing by the

terminator/suspender stating the reasons for early termination or suspension (with the exception of the Sponsor's responsibility for notifying the Regulatory Authorities). After such a decision, the Sponsor and the Principtal vestigator will ensure that adequate consideration is given to the protection of the subjects' interests and safety. The Investigatormust review all subjects as soon as practical and complete all required records.

In addition to the classic assessment of SAEs and the occurrence/severity of other AEs by the Sponsor and then vestigator after exploring potential confounding factors, the following criteria should be considered as guidance for the decision to stop inoculation their subjects:

- A subject experiences an SAE that is related to the inoculum.
- There is insufficient response **©**Z439 and PQP.
- The Investigatorand Sponsor may decide to stop inoculation based on other safety signals not described in the above criteri

# 6 STUDY AGENT

# 6.1 STUDY AGENT(S) AND CONTROL DESCRIPTION

### 6.1.1 ACQUISITION

Challenge Agent(hereafter referred to as inoculum)

# P. falciparum3D7

The P. falciparum 3D7 master cell bankM(CB) was produced from a person with O RM (Negative blood who was infected with the parasite by mosquito bite. The MCB was cryopreserved, aliquoted into cryovials and stored in liquid nitrogen under controlled conditions. Refer to the P. falciparum 3D7 Investigators Brochure for more details [35]. A 3D7 MCB cryovials will be retrieved from storage, thawed, and to aseptically prepare the 3D7 inoculum at Q-Gen.

Study Drug

# <u>OZ439</u>

OZ439 granules+  $\alpha$ -tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension(200 mg and 400 mg strengths of OZ439) will be provided in aluminium sallbets grade sucrose will be provided by Remarm pharmacyThe drug productivil be shipped either directly to QPharm, or via Pharmaceutical Packaging Professionals Pty Ltd (Victoria, Australia). Import will be facilitated by MMV and the TGA will be notifibusing the Clinical Trial Notification (CTN) scheme.

# Piperaquine phosphate (PQP)

Piperaquine phosphate 60 mg will be provided from a stock at Pharmaceutic Backaging Professionals Pty Ltd and hipped directly to Pharm

Antimalarial Rescue Medications

# Riame® andPrimacin<sup>TM</sup> (if required)

Riame® and Primacin will be acquired by QPharm, labelled according to identity, brand or source, and batch number. The supplies will be incompropriate locked storage conditions at Q Pharm until required. The contents of the labelthed rug to be administered to the bjectswill be in accordance with all applicable regulatory requirements. The inoculum Ptradito parum 3D7) used in the challenge model has been proven to be sensitive to the rescue medications.

# Artesunate (if required)

If a subject vomits or cannot tolerate oral drugs, then artesunate will be administered intravenously as described in Section 6.1.5. This drug is the recommended parenteral treatment for malaria in Australia. Currently, it is a Special Access Scheme daung, has been sourced from Guilin Pharmaceutical (Shanghai) Co., Ltd. Import was facilitated by MMV. The manufacture of intravenous (IV) artesunate is undertaken in a WHO-Quelified GMP facility (http://www.mmv.org/access/acces

The rescue drugs, i.e., Rian@etPrimacin<sup>TM</sup>, and artesunate will be inventoried prior to the beginning of trial enrolment on trial accountability loigns regards to condition upon receipt, including lot numbers. Then vestigator or qualified designee will ensure that the received drugs are the specified formulation. The site pharmacist or qualified designee is responsible for maintaining an accurate ientory and accountability record of drug supplies for this trial.

# 6.1.2 FORMULATION, APPEARANCE, PACKAGING, AND LABELING

Inoculum

# P. falciparum3D7

Each 3D7 inoculum dose will contain parasitised and unparasitised RBCs, resuspended in 0.9% Sodium Chloride Intravenous Infusion, in a total volume of 2 mL in syringes. The syringes will be double contained following preparation and labelled in accordant be GCP guidelines and the Access to Unapproved Therapeutic Goodsinical Trials in Australia [44].

# Study Drug

# OZ439

OZ439 is available as  $OZ439 + \alpha$ -tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension dosage form. OZ439 granules TPGS granules are-packaged in a -2 compartment sealed sachet. The OZ439 granules and TPGS granules are physically simparate the sachet packaging. Dose strength &00 mg OZ439 are available. The OZ439 and TPGS granules for oral suspension are mixed with water to form an oral suspension, and sucrose is added prior to administration to the subject. The sucrose is added to make the oral suspension palatable Reconstitution steps will be described in the Pharmacy Maħlualcontents of the label for drug to be administered to the subjects will be in accordance with all applicable regulatory requirements.

# Piperaquine phosphate (PQP)

PQPis formulated as tablets (160g per tablet)PQPwill be labelledaccording to identity, brand or source, and batch number. The contents of the label for drug to be administered to the subjects will be in accordance with all applicable regulatory requirements.

**Antimalarial Rescue Medications** 

#### Riamet®andPrimacin™ and Artesunate

Riame® tablets(20 mg attemether/120 mg lumefantrina) eyellow, round, flat tablets marked with N/C and a score line on one side and CG on the other side. Each carton contains 24 tablets.

Primacin tablets (primaquine phosphate) re round, flat, orange uncoated table imacin tablets are available in bottles of 28 or 56 tab Petismacin will be labelled according to identity, brand or source, and batch number. The contents of the label torug to be administered to the subjects will be in accordance with all applicable regulatory requirements.

Artesunate for I/V administration is presented as a powder for reconstitution (60 mg artesunic acid) in a vial.

#### 6.1.3 PRODUCT STORAGE AND STABILITY

#### Inoculum

#### P. falciparum3D7

The inoculum is prepared at Gen on inoculation day (Day 0). The time between preparation of the 3D7 inoculum and administration to each subject will be a maximum of 2 hours, during which

OZ439 and PQP Protocol Version4.0 QP17C19 27 August2018

time all inocula will be stored on ice. The Renarm pharmacist will downent receipt conditions and time restrictions of use.

Study Drug

#### **OZ439**

OZ439 + TPGS granules for oral suspension drug products should be between 15-30°C. Food grade sucrose to be stored at room temperature.

Piperaquine phosphate (PQP)

PQPtablets are be stored 15 to 25C.

**Antimalarial Rescue Medications** 

#### Riamet®andPrimacir<sup>™</sup>

- Riamet®is to be stored below 30°C and protected from moisture (dispersible tablets).
- Primacin<sup>TM</sup> is to be stored below 25°C.
- Artesunate: store in tightly closed ntainers, protected from light.

All drugs will be held in appropriate locked storage conditions at the clinical unit until required.

### 6.1.4 PREPARATION

Inoculum

#### P. falciparum3D7

The inocula will be prepared asepticallyQ-Gen(QIMR Berghofer), from a frozen cryovial of the P. falciparum3D7 MCB, by nominated QIMR Berghofer staff members under the guidance of the Investigator The infected RBCs will be thawed, washed, resuspended in saline, diluted in a final volume of 2 mL of tinical grade salie, and dispensed into syring [25]. Any remaining unused infected RBCs will be discarded as per approved standard operating procedures.

Study Drug

### **OZ439**

The OZ439 and TPGS granules for oral suspension are mixed with water to form an oral suspensionand sucrose is added prior to administration to the subject. The sucrose is added to make the oral suspension palatable. The will be drunk and then the cup rinse water will be used to swallow the PQP table to reconstitution procedure will be describe the Pharmacy Manual.

# Piperaquine phosphate (PQP)

PQPis available as tablets and no preparation is required tablets will be swallowed with the water that is used to rinse to 2439 suspension cup with.

OZ439 and PQP will be administered at shene tine. Subjects will be fasted for thours preand post-dose.

**Antimalarial Rescue Medications** 

# Riamet®andPrimacin<sup>™</sup>

Riamet®andPrimacir™ are available as tablets and no preparation is required.

#### 6.1.5 DOSING AND ADMINISTRATION

Inoculum

# P. falciparum3D7

An inoculum dose, containing an estimated802 viableP. falciparum3D7 parasitenfected RBCs in a volume of 2 mL, will be administrated intravenously to each subject on Day 0. The actual number of parasites inoculated will take into accountots of viability resulting from cryopreservation, storage and thawing. On inoculation day, subjects may have food until at least half an hour prior to inoculation. Subjects will undergo intravenous cannulation with an appropriate gauge cannula. Placement patency will be checked by flushing the vein with 5 mL of clinical grade saline. The inoculum will be injected, and the cannula again flushed with 5 mL of clinical grade saline. The cannula will then be removed, and haemostasis ensured by use of an appropriate dressing. All subjects will be inoculated intravenously within 60 minutes of each other. See Section 6.1.3 for stability informatiAn. extra syringe will be prepared to quantify the parasite count of the inocula by malaria 18S qPCR.

### Study Drug

# OZ439and piperaquine phosphate (PQP)

Subjects will be admitted to the clinical unit fixingle dose administration £672439 and PQP8 days after malaria inoculation earlier if a subject has amalaria clinical score >60r at Investigators discretion. The doses to be administered to subjects in Cohrantd12areshown in Tables 1 and 2 respectively(Section 4.1.) Subsequent doses for subsequent cohorts will be determined by the LEGRT following safety tolerability and PK/PD review. Subjects will be fasted for ≥6 hours pre and pos£72439 and PQPadministration. The OZ439 TPGS granules will be mixed with water to form a suspension. Sucrose will be added to the suspension to assist with palatability. PQP tablets will be administered in the suspension and swallowed

with the OZ439 cup rinse water he reconstitution procedure will be described in the Pharmacy Manual.

**Antimalarial Rescue Medications** 

# Riame® andPrimacin™

All subjects will receive compulsory treatment Riamet® on trial Day42±2, or at failure of OZ439 and PQP to clear parasitaemia, or at evidence of recrude to the description of stage parasites/mL and to description and to description and the description of the line and the description of the line and the description of the line and the description of the line and the description of the line and

Subjects may also be treated hwPrimacin at the time of Riam treatment gametocytaemia is suspected from parasite lifecycle stage transfer or by the presence of stable low level parasitaemia, or at the vestigators discretion, to ensure complete clearance of gametocytes. If needed, subjects will take 6 Primatentablets, each containing 13.2 mg primaquine phosphate equivalent to 7.5 mg primaquine (the total primaquine dose will be 45 mg). Primater use will be taken as single dose with food. Subjects will be reminded of the potential side effects of Primacin and given the Consumer Medicine Information for Primate (Appendix 1)

IV artesunate may be used as a rescue medidationubject vomits or cannot tolerateal drugs. See artesunate section above.

### 6.1.6 ROUTE OF ADMINISTRATION

Inoculum

P. falciparum3D7

Intravenous

Study Drug

Artefenomel (OZ439)

Oral administration

Piperaguine phosphate (PQP)

Oral administration

**Antimalarial Rescue Medications** 

Riamet®andPrimacin™

Oral administration

#### Artesunate

If a subject vomits or cannot tolerate oral drugs, then artesunate will be administered intravenously as described in Section 6.1.5.

### 6.1.7 STARTING DOSE AND DOSE ESCALATION SCHEDULE

Dosing with the malarianoculumand rescue drugs is presented in Section 6.1.5. No dose escalation will be performed.

# Study Drug

Dosing with OZ439 and PQWill be performed as described in section 4.1. The doses of OZ439 and PQP for subjects enrolled in cohort 1 are shownable 1 of the Protocol Summa Syubjects will be randomised to one of the four groups that comprise Cohort doses of OZ439 and PQP for subjects enrolled in cohort 2 are shown in Table 2 of the Protocol Sum South jects will be randomised to one of the two poups that comprise Cohort The OZ439 and PQP doses to be evaluated is ubsequent cohortwill be determined at the SDRT meetings bed on the afety and tolerability data up to Day42±2, and PK/PD analysis outcomes (based on PD data up to Day42±2 and PK data up to Day435±2) of the drugs given in combination previous Cohort(s).

The doses used in all Cohorts will not exceed 800 mg for OZ439 and 1440 mg for PQP as determined in previous safety, pilot efficacy and phase 2 studies.

### 6.1.8 DOSE ADJUSTMENTS/MODFICATIONS/DELAYS

Not applicable.

#### 6.1.9 DURATION OF THERAPY

See Seioon 6.1.5 for dose information.

#### 6.1.10 TRACKING OF DOSE

The P. falciparum challenge agent, OZ439 and PQAnd if requiredPrimacin™ will be administered at the clinical unit the presence of clinical unit staff. Subjects may be administered

Riamet®on site for initial dosing followed by moitoring, either in the clinicor by phone for 3 days to ensure adherenceRiamet®therapy.

#### 6.2 STUDY AGENT ACCOUNTABILITY PROCEDURES

The QPharm pharmacist or delegate, as nominated by the Prinhorized tigator is responsible for maintaining accurate study agent accountability records throughout the study. Study agents include the challenge agents (OZ439 and PQP), and the rescue medications. Dispensing, accountability and documentation will be in accordance with Pharm standard procedures. All products will be inventoried upon receipt by the Poarm pharmacist. The condition of the products at the time of receipt by the pharmacist will be documented, as will the time restrictions of use for the syringes containing the challenge agents of the time restrictions of use for the oral suspension of OZ439 and TPGS The lot numbers and expiry dates of the inoculum and antimalarial drugs will be documented. The oarm pharmacist or delegate will ensure that the received products are the specified formulation.

The storage, handling and the disposal of the challenge agents will be in accordance with approved procedures. All dosages prescribed and dispensed to the subjects and all dose changes during the study must be recreded in the eCRF. It drug supplies are to be used only in accordance with this protocol, and not for any other purpo. It used medications will be fully document. It does not unused drug containers must be destroyed at the site once drug accountability and has been checked by the Sponsor or its delegate, and written permission for destruction has been obtained from the Sponsor.

Study products and study accountability logs will be available to the Sponsor or their representative as part of thecesy monitoring procedures. Upon completion of the study, copies of all study drug management records will be provided to the Sponsor. Original records will be maintained at the clinical site with the rest of the study records.

### 7 STUDY PROCEDURES AND SCHEDULE

# 7.1 STUDY PROCEDURES/EVAUATIONS

#### 7.1.1 STUDY SPECIFIC PROCBURES

# Medical history

Medical history will be elicited at screening as described below.

| Past Medi | cal/Surgi | cal Histo | ry Inc | ludes: |
|-----------|-----------|-----------|--------|--------|
|-----------|-----------|-----------|--------|--------|

History of all known allergies

Current medications, including overecounter and herbal preparations

| listory of substance abuse and recreational drug use | |
|---|---|
| listory of depression, anxiety, mental illness, emotional problems, use of psychiatric m | nedication |
| Surgical procedures and results | |

#### Physical examination

# Complete Physical Examination Includes:

| Weight(Screening only) |
|---|
| Height (Screening only) |
| Review of systems excluding genitourinary examination and including the following: |
| Head, neck (including thyroid), ears, eyes, nose and throat |
| Heart/circulation |
| Chest |
| Lungs |
| Abdomen |
| Skin |
| Neurological exam |

Abbreviated Physical Examination abbreviated physical examination will be performed at Day 0 (inoculation day) and Day 8 (OZ439/PQP dosing day). The examination will include; heart/circulation, chest, lungs and abdomen.

SymptomDirected Physical Examinationphysical examinations will be symptomirected at specifiedtime points Body systems will be reviewed only if clinically indicated at the discretion of the Investigator (see Appendix for a list of symptoms and signs of malaria)

### Beck Depression Inventy

All subjects will be required to complete the Beck Depression Inventory at screening. This is a validated questionnaire used as an objective tool for the assessment of depression (See Appendix 4).

# Vital signs/12lead ECG and Safety Laboratory Samblewed Time Windows

| Time point Tolerance window | |
|----------------------------------------------------------------|----------|
| Vital Signs/ 12Lead Electrocardiogram/Safety Laboratory Sample | |
| In conf | finement |
| Predose - 90 min to 0 h | |
| 0-4 hours inclusive after IMP | ± 10 min |
| 4-12 hours inclusive after IMP | ± 10 min |
| 16-72 hoursinclusive after IMP ± 40 min | |
| Out patient | |

| 72-120 hours inclusive | ± 120 min |
|------------------------|------------|
| 168-EOSinclusive | ± 48 hours |

# Vital signs

Vital signs (temperature, heart rate, respiratory rate and blood pressure) will be measured at screening after the subject has rested in the supine position for at least 5 minutes and in the standing position within 23 minutes when changing from the supplies standing position (blood pressure and heart rate only). At all other timperints, vital signs will be measured after the subject has rested in the seated position for at least 5 minutes. Tympanic temperature will be taken at the clinical unit

The normal ranges for vitalignsonce on study are:

| Parameter | Range |
|--------------------------|-------------------|
| Systolic blood pressure | 90-140 mmHg |
| Diastolic blood pressure | 50-90 mmHg |
| Heart rate | 50-100 bpm |
| Temperature | 35.037.5°C |
| Respiratory rate | 10-25 breaths/min |
| Peripheral O2 Saturation | >=95% |

# Electrocardiograms

Triplicate 12lead ECG will be recorded after restingsupine for at least fininutes The same body position will be assumed by the subject for each recording. ECG tracings will be retained and labelled as per standard procedures at the and the mean of the three values will be recorded in the eCRFAny clinically, significant indings will be discussed with the Medical Monitor and Sponsor and documented as adverse events. The Investigator will sign and date each ECG as evidence of their review.

The normalECG rangesonce on study are:

| Parameter | Range |
|-------------|---------------------|
| PR interval | <= to 210 ms |
| QRS | >50 to < = to120 ms |
| QT interval | >200 to < 500 |
| QTcB/QTcF | Males: ≤ 450 msec |
| QTcB/QTcF | Females ≤470 msec |

# **Blood sampling**

Main Study Blood will be collected for clinical labatory evaluations including haematology, biochemistry serology, pregnancy testing nd or FSH testing (see Section 7.2.1). Blood samples will also be collected to monitor malaria parasitaemia and to quantify plasma outrogentrations for PK analysis (see Section 7.2.2).

Optional exploratory components Blood will be collected to characterise specific cell subsets with an aim to identify immune regulatory pathways initiated during malaria infection that can be targeted for clinical advantage. Blood samples will also be collected to investigate early changes to RBC that leads to malaria induced anaemia.

The estimated blood volume required **both** the main study and optional exploratory components is listed in Appendix2. The total volume of blood drawn from each subject will not exceed 450 mL in any given 30day period The total blood volumet day 30 for both the main study and optional exploratory components, will be approximately 40 and and optional exploratory components, will be approximately 40 and optional exploratory components, will be approximately 40 and optional exploratory components.

This volume provides an allowance for unscheduled safety laboratory assessments that may be required at the discretion of the Principal vestigator the Sponsor to ensure subject safety.

# Urine sample collection

Urine will be collected for urinalysis and drug screening (Seetion 7.2.1).

# AE recording

AEs will be recorded as described Section 8.

#### Malaria Clinical Score

The following 14 signs/symptoms frequently associated with malaria will be glaydiaded. Study nurse ordoctorusing a 4point scale (absent; 6nild: 1; moderate: 2; severe: 3) and summed to generate a total Malaria Clinical Score (maximum score possible is 42). Individual scores for each symptom as well asset total score will be recorded

| Headache | Anorexia |
|-----------------------------------------|----------------------|
| Myalgia (muscle ache) | Nausea |
| Arthralgia (joint ache) | Vomiting |
| Fatigue/lethargy | Abdominal discomfort |
| Malaise (general discomfort/uneasiness) | Fever |
| Chills/Shivering/Rigors | Tachycardia |
| Sweating/hot spells | Hypotension |

#### **Medical Diary**

Provide subjects with diary cards and instraubjects to record symptoms and concomitant medications during the study.

Temperature Self Recording

Provide subjects with thermometers to record any temperature readings during the study in the event of symptoms of fevesublingual temperature will **te**ken by subjects at home for practical reasons.

### 7.1.2 STANDARD OF CARE STUDY PROCEDURES

Not applicable.

#### 7.2 LABORATORY PROCEDURES/EVALUATIONS

### 7.2.1 CLINICAL LABORATORY EVALUATIONS

Any significant deviations from results obtained during screening will bllowed until resolution or investigated fully, or until the subject is referred to a general practitione in westigator will document the clinical significance of all results falling outside of the normal reference ranges. All abnormal laborator test results judged as being clinically significant will be record to the normal reference ranges.

The estimated blood volume required for these tests is listed in Appendix

# <u>Haematology</u>

| Full blood count (FBC) with differential |
|---|
| White blood cell count (WBC) |
| WBC differential (diff) |
| A manual blood smear should be reviewed if there are immature/abnormal cells detected |
| automated differential or if an automated differential was not able to be performed. |
| Neutrophils (NEUT) |
| Lymphocytes (LYM) |
| Monocytes(MON) |
| Eosinophils (EOS) |
| Basophils (BAS) |
| Red blood cell count (RBC) |
| Mean corpuscular volume (MCV) |
| Haemoglobin (HGB) |
| Haematocrit (HCT) |
| Platelet count (PLAT) |
| Reticulocyte count (RETI(screening and EOS or early termination visit only) |
| Blood Group and Rh(D) tes(Screening only) |

# **RBC** alloantibodies testing

Blood for RBC alloantibodies testing will be collected at screening Date 45±2 or early termination visit.

# **G6PD** testing

Blood for G6PDtestingwill be collected at screening on 6PDdeficiency is not an exclusion criterion but will be determined at screening to ensure the safety of Primacin<sup>TM</sup>.

# Coagulationtesting

Blood for PT, APTT and INR will be collectealt screening visit.

# Biochemistryand CRP biomarker

| Sodium (SODIUM) | Alkaline phosphatase (ALP) |
|---|---|
| Potassium (K) | Alanine aminotransferase (ALT, SGPT) |
| Chloride (CL) | Aspartate aminotransferase (AST, SGOT) |
| Bicarbonate (BICARB) | Calcium corrected |
| Glucose (GLUC) | Phosphate (PHOS) |
| Urea | Lactate dehydrogenase (LDH) |
| Creatinine (CREAT) | Magnesium(Screening only) |
| Urate | Cholestero(Screening only) |
| Albumin (ALB) | Triglycerides(Screening only) |
| Globulin | HDL (Screening only) |
| Total protein | Estimated glomerular filtration rate (eGFR |
| Total bilirubin (BILI) | C-Reactive Protein (CRP()Not included at |
| | Screening |
| Direct (conjugated) bilirubin (BILDIR) | |

### Urinalysis

Urine will be tested by dipstick at the clinical unit. If there are any abnormalities considered clinically significant in blood, leucocytes or protein, the urine will be sentonical laboratory urinallysis per the clinical unitandard procedure.

| Glucose (GLUC) |
|---------------------------|
| Bilirubin (BILI) |
| Ketone (KETONES) |
| Specific gravity (SPGRAV) |
| Blood |
| рН |
| Protein (PROT) |

| Urobilinogen (UROBIL) |
|-----------------------------------------|
| Nitrite |
| Leukocytes (WBC) |
| Formal laboratory urinalysisf required) |

# Urine drug screens and alcohol breath tests

If the results of the urine drug screens or alcohol breath tests are positive, subligates be enrolled in the clinical study

All subjects will be questioned bout concomitant medications and use of recreational drugs. The urine drug screen may be repeated if the potential subject denies usage of any of these agents and the test result is believed to be a false positive.

Subjects testing positive for paracetamol at screening and/or inoculation day may still be eligible for study participation, at the vestigators discretion. Subjects requiring paracetamol on a daily basis would not be eligible to enrol in the study, has use of any overhe-counter medication during the study is restricted and potential subjects should not discontinue their usual medications in order to participate in the study.

| Urine drug screens: | |
|---------------------|---------------------------------|
| Amphetamines | Opiates |
| Methamphetamines | Phencyclidine |
| Barbiturates | Tetrahydrocannabinol (cannabis) |
| Benzodiazepines | Tricyclic antidepressants |
| Cocaine | Acetaminophen (paracetamol) |
| Methadone | |
| Alcohol breath test | · |

# Serology

| HIV 1/2 (anti-HIV1 and antiHIV2 Ab) |
|---|
| Hepatitis B (HBs Ag, antHBc (IgG + IgM if IgG is positive)) |
| Hepatitis C (antHCV) |
| Hepatitis A (antiHAV) (IgM) - performed from stored sample for testing, attvestigator's discretion |
| Hepatitis E (antHEV) (IgM) - performed from stored sample for testing, and the stigator's discretion |
| EpsteinBarr virus- performedfrom stored sample for testing, and the stigator's discretion |
| Cytomegalovirus performed from stored sample for testing, attvestigator's discretion |

# Safety serum storage

Blood for serum storage as safety retention sampiles collected at times outlined in Section 7.3.

### 7.2.2 OTHER ASSAYS OR PROEDURES

The estimated blood volume required for these tests is listedpendix2.

### PK/PD AllowedTime Windows

| Time point | Tolerance window |
|---------------------------------|------------------|
| Pharmacokinetic/pharmacodynamic | |
| In confinement | |
| Predose | - 60 min to 0 h |
| 0-4 hours inclusive after IMP | ± 2 min |
| 4-12 hours inclusive after IMP | ± 5 min |
| 16-72 hours inclusive after IMP | ± 30 min |
| Out patient | |
| 72-120 hours inclusive | ± 120 min |
| 168EOS | ± 48 hours |

### Malaria monitoring

Blood will be collected to monitor parasitaemia using Cor targeting the 18S rRNA gene. Additional blood (up to approximately 2.5 mL per timpeint) may be collected for parasite lifecycle stage qR-PCR at thenvestigators discretion. This is to evaluate for the presence of sexual parasite stages (gametocytes) and other parasite lifecycle stages in the blood. This blood may also be used for research into various aspects of parasite biology e.g. gametocytes, parasite lifecycle stages, excrudescence, commitment etc. The qROR may target genes including but not limited to: the female gametocytepecific transcriptofs25, the male gametocytespecific transcriptofMGET, and the ringstagetranscriptofSBP1 as appropriate. The samples not return at time points indicated by malaria 18S qPC-Br, at the Investigator's discretion.

Microscopic examination for evidence of parasitaemia or gametocytaemia may be conducted at the Investigator's discretion.

Malaria monitoring will continue until aninimum of onenegative 18 qPCR is detected post rescue therapy

# PK blood collection and processing

Blood sampling for PK analysis will be performed at scheduled time provints immediately before dosing with OZ439and PQP until 816 hours postdose, (allowed timewindows as described abov)e

Blood samples will be collected either by direct epuncturer via an indwelling cannula inserted in a forearm vein. Details of the volume of blood collected are listed in Appendix 2.

A description of the required laprocedures will be described in the Laboratory Manual.

The actual sample collection date and time will be entered in the PK blood collection section of the eCRF. Any sampling problems will be documented in the eCRFs.

# Pharmacokinetianalytical methods

Plasma concentrations of OZ439 and R@Pbe quantified by LC MS/MS in the selected reaction monitoring mode using heated electrospranjzietion in positive ion mode.

OZ439: Plasma samples will be precipitated with five volume equivalents of a mixture of acetonitrile/methanol (4/1, v/v) containing the internal standard. After centrifugation, the samples will be diluted with a mixture of water/acetonitrile (1/1, v/v). An aliquot of 2  $\mu$ L of the sample be injected onto the ligh-performance liquid chromatographystem (HPLC).

PQP. Plasma samplewill be precipitated with ten volume equivalents of acetonitrile containing the internal standard. After centrifugation and dilution with one equivalent ter, an aliquot of 25.0 µL of the supernatamill be injected onto the HPLC system.

# Optional exploratory components

Blood sampling formmune cell characterisation and complement regulatory protectives will be performed at scheduled time points detailed in Section 7.3. The time into for the exploratory components rescheduled to coincide with blood collection time into of the main study. If timepoints of the main study change the exploratory study-time will change to match to ensue subject comfort and convenience.

Blood samples will be collected either by direct venepuncture or via an indwelling cannula inserted in a forearm vein. Details of the volume of blood collected are listed in Appendix 2.

#### Optional exploratory components alytical methods

Specific cell subsets will be sorted from blood collected by so (prior to malaria inoculation) 4, 8(prior to OZ439 and PQP administration 5 and at EOS. The host immune response generated by these sorted cells will be investigated the DNA, RNA and protein levels with an integrative high dimensional multiomics strategy. DNA, RNAs, including mRNA, microRNA and lenger coding RNA (IncRNA), and proteins will be extracted from the same sample and samples will be assayed in a highimensional biology approach. mRNA, miRNAs, and IncRNA will be profiled using NanoString, RNAseq, and/or whole transcriptome analysis. Comprehensive panels of molecules involved in T cell activation, function, and exhaustion will be evaluated using multi parametric flow cytometry. Proteogenomics will also be investigated, whereby data from high resolution masspectrometers (e.g. QTRAP) will generate fingerprints for peptides which are mapped against NGS transcriptomic and genomic data

Expression of complement regulatory proteins (CD35, CD55, and CD59) and phosphatidylserine on RBC will be assessed by flow cytometanyd will be quantified by commercial ELISArom blood samples collected n Day 0(prior to malaria inoculation), Day (prior to OZ439 and PQP administration), Days 10, 12, 13, 15, 18 and at EOS.

# 7.2.3 SPECIMEN PREPARATION HANDLING, AND STORAGE

Q-Pharm's standard work instructions will apply to the allowed time windows for study procedures and sample collection. If the observation time and blood sampling time coincide, for precision of timing, blood collection will take precedence over other **pduc**es scheduled at the same time.

Blood will be collected into tubesontaining the appropriate actingulant. Samples will be processed according to the laboratory requirements.

Biological samples will be retained for the time required for assessmentabysis, and may then be discarded. Safety serum samples will be stored indefinitely with the permission of the subjects for any retrospective safety assessments.

### 7.2.4 SPECIMEN SHIPMENT

Samples collected will be shipped to nominated local or intermattlaboratories for assessment (Section 1) The site staff will be responsible for shipment of samples to analytical laboratories for testing. Samples must be packed securely together with completed shipment forms in shipping containers together with the time of the samples

#### 7.3 STUDY SCHEDULE

#### 7.3.1 SCREENING

A screening visit will be schedulædter an initial phone interview conducted by clinical unit staff has occurred to review background information. For the screening visit, potential subjects will be asked to come to the clinical unit after an overnight fast of ≥8 hours. During this initial screening visit, anInvestigatowill discuss the details of the study wtthe potential subjectand the potential subject to ask questions.

Individuals willing to be considered for inclusion may sign the Consent Form during the screening visit, or return to the clinical unafter further consideration. The subject will be given a copy of the Participant Information Sheet and signed Consent Form for their records. The signed and dated

originals will be held on file by the clinical unlaticipation consent must be obtained all subjects prior to screening tests.

The consenting process will take place with one of the arm medical staff denvestigatos and will include the following:

- 1. Provide the Partipation Information Sheet and formed Consent Form and give the subject sufficient time to review the contents.
- 2. Explain the study via the Participation Information Sheet and gain informed consent from the subjectif they are willing to consent.
- 3. Ensure the subjected member of staff taking consent havened and detailed the Informed Consent Form and received a signed copy.

Once the potential subject has provided written consent to participate, the dyscreening may be initiated. The screening will be conducted within 4 weeks prior to the inoculation day and will include:

- 1. A screening number will be assigned to each subject.
- 2. Elicit a complete medical history and use of medications.
- 3. Elicit a social history includingecreationaldrug, alcohol and tobacco use.
- 4. Perform alcohol breath test.
- 5. Perform a drugs of abusereen.
- 6. Perform complete physical examination.
- 7. Ask subject to complete the Beck Depression Inventory.
- 8. Assess the cardiovascular disease risk as per exclusion criterion 4.
- 9. Record vital signs.
- 10. Obtain a 12ead ECGn triplicate
- 11. Collect urine for urinalyssi.
- 12. Collect blood samples for haematology, biochemistry, RBC alloantibodies, G6PD testing, and serology (viral hepatitis B and C and HIV).
- 13. Collect blood for coagulation profile
- 14. Perform serum β-hCG pregnancy test for all female subjects and follicle stiting hormone test(FSH) for postmenopausal females.
- 15. Verify subject meets inclusion/exclusion criteria.

Subjects who complete all screening procedures and satisfy all entry criteria will be considered eligible to participate in this study. To be eligible future future, laboratory values at screening must not be outside the range of the normal values at a level deemed to be clinically significant according to Sponsærpproved criteriaFor eligibility parameter, a repeat may be requested exclude laboratory error. Recreening will not be allowed unless three vestigator considers the cause of the initial precreening failure to be of an acute and completely reversible nature.

If screening laboratory results are abnormal, e.g. HIV testing, the subject will be referred for appropriate counselling. If any clinically significant abnormalities are detected during screening, the subject will be referred for follows tests to a genear practitioner or medical specialist as appropriate.

### 7.3.2 ELIGIBILITY CONFIRMATION VISIT

Day -3 to Day -1 safety visit

Subjects (including approximately 4 reserve subjects s mentioned in Section 5.4 will report to the clinical unit between Day3 to Day-1 for the following baseline assessments, unless screening laboratory assessments were conducted within this period, in which case repeat sampling will not be required.

This visit will include:

- 1. Collect blood samples for haematologyjochemistry (including CRP biomarke) and serum β-hCG pregnancy test for all female subjects
- 2. Collect urine for urinalysis.

The timing of these assessments is to ensure that results are available for revidwhesting to prior to inoculation or inoculation day Subjects with clinically significant laboratory findings at this stage will not be eligible for inoculation.

Malaria inoculation day (Day 0)

Each subject (analoproximately4 reservesubjects) will report to the linical unit on the morning of Day 0. The Investigator will review the subjects' screening and eligibility confirmation visit results prior to their enrolment into the stuadyd subsequent inoculation he Investigator will emphasise the requirement to retutto the dinical unit for malaria drug treatment the malaria inoculation and confirm that they will not be living alone from Day 0 until the end of the study by checking housemates contact details recorded at screening visit.

On admission to the linical unit, subjects will be required to undertake further procedures to determine whether they remain eligible to be enrolled. A reserve subject may be asked to replace a subject who does not continue to meet eligibility. These reserves will be compensated for the study visit even if not inoculated, as described in the Participant Information and Consent Form.

The procedures that will be undertaken prior to inoculation Day Oinclude:

- 1. Verify that all applicable eligibility criteria have been met.
- Elicit information regarding any new medical conditionidinesses and medication use since screening.
- 3. Perform alcohol breath tested urine drug screen
- 4. Perform urine β-hCG pregnancy test foll/OCBP subjects

- 5. Conductabbreviate physical examination
- 6. Record vital signs.
- 7. Obtain 12lead ECGn triplicate.
- 8. Cannulate subjects with an indwelling intravenous cannula for the malaria inoculum, and record which arm is utilised.
- 9. Collect blood samples for malaria qPCR and safety serum storage.
- 10. Collect optional blood samples for immune cell characterisation and complement regulatory proteins (if consented separately).
- 11. Perform Malaria Clinical Score.

### Administration of the malaria inoculum:

- 1. Administer the malaria inoculum of \$200 viable P. falciparum 3D7 infected human RBCsintravenously in the morning (approximately 9:00 AM).
- 2. Observe for a minimum of 60 minutes after inoculation to evaluate for immediate adverse reactions.
- 3. Educate subjects on signs and symptoms of malaria (App®)ndix
- 4. Emphasise to subjects the importance of returning on the nominated day (approximately Day 8), or as advised by the clinical unit staff, **MaP** antimalarial treatment.
- 5. Provide subjects with diary cards and thermometers to record any temperature readings during the study in the event of symptoms of fever. Subjects will also record symptoms and concomitant medications on the diary cards during the study.
- 6. RecordAEs and concomitant medications.
- 7. Record vital signs prior to leaving the clinical unit (approximate) a 60 minutes after inoculation).
- 8. Record malaria clinical score prior to leaving the clinical unit (malaria clinical score baseline sample; see Section 7.1.1).

#### 7.3.3 FOLLOW-UP

Malaria monitoring via phone (Days 13)

During this period, subjects are exped to be asymptomatic. A daily phone call or text message will be made to the subjects by clinical unit staff to monitor subject by and to solicit any AEs.

Daily visits to the clinical unit for malaria monitoring (Day 4 AM until qPCR positive for malaria)

Follow-up from Day 4 until qPCR becomes positive will be undertaken through daily visits (approximately 8:00 AM) to the clinical site.

The following procedures will occur during these txisi

- 1. Performsymptom-directed physical examination on signs or symptoms of malaria are identified and it is clinically indicated (Appendix).
- 2. Elicit information regardig any new medical condition in the since screening
- 3. Record vital signs.
- 4. Collect blood sample for malaria 18S qPCR.
- 5. Collect optional blood samples for immune cell characterisation, Day & separately).
- 6. Record malaria clinical score.
- 7. RecordAEs and use of concomitant medications.
- 8. Check subjectiaries.

Day when qPCR positive until treatment day (Day 8)

Follow-up from the day that malaria 18S qPCR becomes positive until treatment day will be undertaken through twice daily (AM & PM) visits to the clinical site separated by approximately 12 hous (i.e. 06:00- 11:00 and 18:00 23:00). The following procedures will occur during these visits:

- 1. Performsymptom-directed physical examination
- 2. Elicit information regardig any new medical condition in the since screening
- 3. Record vital signs.
- Collect blood sample for malaria 18S qPCR.
- 5. Record malaria clinical score.
- 6. RecordAEs and use of concomitant medications.
- 7. Check subject diaries.

In-patient observation and IMP antimalarial treatment phase (Day8-Day 11) Subjects will be admitted to the clinical unit for 2 hourson the morning of Day8 (or earlier if a subject has a malaria clinical score >6 or at Investigator discretion) for OZ439 and PQP treatment and monitoring of clinical symptoms of malaria.

# Admission

The following procedures will occur at admissiontheclinical unit:

- 1. Performabbreviate only sical examination
- 2. Perform alcohol breath tested drug screen
- 3. Elicit information regarding any new medicanditions or illnesses.

- 4. Record vital signs.
- 5. Obtain12-lead ECGn triplicate.
- 6. Collect urine for urinalysis.
- 7. Perform urine β-hCG pregnancy test foll/OCBPsubjects
- 8. Cannulate subjects with an indwelling intravenous cannula.
- 9. Collect blood samples for aematology, biochemist (including CRPbiomarke), malaria 18S qPCR (parasite clearance baseline sample), and PK analysis (measur @ 2489 of and PQRevels; PK baseline sample).

NOTE: As these test results may not be available before the drug adationis, the results of this time point will be used for future interpretation of study results.

- 10. Collect optional blood sample for immune cell characterisation and complement regulatory protein (if consented separately)
- 11. Record malaria clinical score.
- 12. Record AEs and use of concomitant medications.

# Treatment and observation

The following procedures will occur during treatment and observation:

- Administer the appropriate doses of OZ439 and PQP to fastedours)subjectsunder direct observationasdescribed in (Section 6.1.5)
- 2. Follow up subjects as inatients for 72 hours to onitor safety and tolerability the treatment and adequate clinical response.
- 3. Performsymptom-directed physical examination when signs or symptoms of malaria are identified and it is clinically indicated.
- 4. Obtain12-lead ECG irtriplicate at 4, 6, 8, 1224 and 72 (D4) hours postOZ439 and PQP administration
- 5. Record vital signs 3 times a day whilst confined.
- 6. Record malaria clinical score 3 times a day whilst confined.
- 7. Collect blood samples for malaria 18S qPCR following treatment 4at8, 12, 16, 20, 24, 30, 36,42,48, 60, and 72 hours per 2439 and PQP administrations per allowed time windows
- 8. Collect blood samples for PK analysis@Z439andPQPat 0.5, 1, 2,3, 4, 5, 6, 8, 12, 16, 24, 48, and 72 hours pe@Z439 and PQPadministration as per allowed time windows
- Collect optional blood samplesfor complement regulatory protein(if consented separately) approximately 48 ourspost OZ439 and PQP treatment.
- 10. RecordAEs and use of concomitant medications.

#### Prior to exit from the clinical unit

Subjects will be allowed to leave the clinical unit 72 hquostOZ439 and PQPreatment at the Investigators discretion.

The following procedues will occur prior to discharge from the clinical unit:

- 1. Performsymptom-directed physical examination Investigators discretion
- 2. Record vital signs.
- 3. Collect blood samples for haematology, biochemistimus luding CRP biomarke), PK analysisandmalaria 18S qPCR-72hourspostOZ439 and PQPdosing).
- 4. Obtain 12lead ECG in triplicate
- RecordAEs and use of concomitant medications.

Out-patient monitoring post-OZ439 and PQPtreatment (Day 12 up to Day42±2)

Follow-up at either AM (approximately 08:00) or AM and PM (if necessary, approximately 12 hours apart) will be undertaken on an-patient basis through visits postinfinement for clinical evaluation and blood sampling.

The following procedures will tackplace during these visits:

- 1. Elicit information regarding any new medical conditions or illnesses.
- 2. Collect a blood sample for malaria 18S qPi@Rhemorning andn the evening on days 12 and 13 and thethree times weeklip at Investigatos discretion based or parasitaemia until Day 42±2.
- 3. Collect blood samples for parasite lifecycle stage **GRCIR** at thenvestigators discretion (Section 7.2.2).
- 4. Collect blood samples for PK analysis of OZ439 and PQP £2,9668±48, 240±48, 336±48, 504±48, 672±48 and 840±48 hoursafter OZ439 and PQP administration.
- 5. Collect blood samples for haematology and biochem (strc/) uding CRPbiomarke) and urine for urinalysis at 336±48, 504±48 and 672±48 hours postOZ439 and PQP administration at the Investigator's discretion.
- 6. Collect optional blood samples for complement regulatory proteinsconsented separately at 96±2, 120±48, 168±48, 240±48 hourspostOZ439 and PQP
- 7. Collect optional blood samples formune cell characterisation consented separately) at 168±48 hourspostOZ439 and QP.
- 8. Performsymptom-directed physical examination of signs or symptoms of malaria are identified and it is clinically indicated.
- 9. Record vital signs.
- 10. Record malaria clinical score if vital signs are abnormal or anthestigators discretion.
- 11. RecordAEs and use of concomitant medications.
- 12. Check subject diaries.

All subjects will receive a standard course of therapy Rithmet® (artemethelumefantrine) on trial Day 42±2 or earlier in the event of failure of clearar or ecrudescence of parasitae ror i at Investigators discretion based on subject safety.

- Failure of clearancedefined asailure to clear parasitaemia by at leastfolio at 72 hours postIMP administration
- Recrudescence: defined <u>a</u>\$ 000 blood stage parasites/mL and a 2-fold parasitaemia increase within 48 hours, or-occurrence of malaria symptoms with a mialaclinical score >6.)

Subjects may take the doses at the clinical **ornia**t home, as determined by **threv**estigator Subjects will receive a phone call or text message from clinical unit staff to check on symptoms and ensure compliance and completion of treatment following the doses taken at the time of Rianue tatment (Setion 6.1.5).

The following procedures will be performed priorRoame® treatment

- 1. Elicit information regarding any new medical conditions or illnesses.
- 2. Perform symptomdirected physical examination.
- 3. Record vital signs.
- 4. Collect blood samples for haematoly, biochemistry including CRP biomarke).
- 5. Collect blood samples formalaria 18S qPCR, and parasite lifecycle stapser-PCR (if required).
- 6. Collect blood samples for PK analysis of OZ439 and PiQRiamet®treatment occurentrial Day42±2.
- 7. Record malaria clinical score if vital signs are abnormal or athtrestigators discretion.
- 8. RecordAEs and use of concomitant medications.
- 9. Obtain 12lead ECGn triplicate.
- 10. Check subject diaries.

Follow-up post rescue treatment Riamet is administered prior to Day 42±2

For all subjects a followup visit will occur 3days(+2-days)after initiation of Riamet treatment The following procedures will be performed this visit.

- 1. Perform symptom directed physical examination.
- 2. Record vitalsigns.
- 3. Collect blood samples for haematology, biochemi@trogluding CRPbiomarke).
- 4. Collect blood formalaria 18SqPCR (if the result is positive the subject will be followed up until a minimum of one negative qPCR is detected).

The following procedures will be performed the EOS visitafter completion of Riame treatment (Day 45±2):

- 1. Elicit information regarding any new medical conditions or illnesses.
- 2. Performfull physical examination.
- Record vital signs.
- 4. Collect blood samples for haematology, biochemistroluding CRPbiomarke),
- 5. Collect blood formalaria 18SqPCR(if the result is positive the subject will be followed up until a minimum ofonenegative qPCRs detected).
- 6. Collect blood forparasite lifecycle stageRT-PCR (if required).
- 7. Collect urine for urinalysis
- 8. Record malaria clinical score
- 9. Collect blood samples for RBC alloantibodieerologyand safety serum storage (2 serum samples).
- 10. Collectoptional blood samples immune cell characterisation complement regulatory proteins (if consented separately).
- 11. Performserumβ-hCG pregnancy test foll/OCBPsubjects
- 12. RecordAEs and use of oncomitant medications.
- 13. Obtain 12lead ECGn triplicate.

See Section 8.3 for follows procedures for ongoing AEs/SAEs.

#### 7.3.5 EARLY TERMINATION VISIT

If withdrawal occurs at any stage of the study, the subject will be **asked**mplete an EOS evaluation. In addition, subjects are informed of the essential requirement to complete the antimalarial drug treatment for their safety, via the Participant Information Sheet.

Participation in an early termination evaluation by each is voluntary. Procedures during the early termination visit are the same as for the 45 and EOS visit (Section 7.3.4).

#### 7.3.6 UNSCHEDULED VISIT

Unscheduled visits for malaria 18S qPCR or safety monitoring may be required at the Investigators discretion based on parasitaemia, clinical symptoms or laboratory results. Subjects will be contacted by phone to arrange these visits. Where possible, visits will be arranged at a time that is both convenient for the subject and meets any clinical urgencyters ided by the Investigator Unscheduled visits will be documented in the source documents and eCRF.

#### 7.3.7 SCHEDULE OF EVENTS TABLE

The Schedule of Events Table summarises the procedures to be conducted as per this protocol during screening, confinement a postconfinement. Section 7.1 and 7.2 provide detailed information on the procedures.

An experienced nurse will be in attendance at the clinical which subjects are exite and the Investigator will be available within approximately 30 minutes call back if required.

In the schedule of events, evaluation may be in the morning, between 6:00 AM to 11:00 AM, and in the afternoon, between 6:00 PM to 11:00 PM, therefore separated by approximately \$12\$

Some safety and laboratory evaluation days may vary ±2 days based on qPCR counts and clinical unit visits at thenvestigators discretion.

Table 2: Schedule of Events

| Table 2: Schedule of Events | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Screening<br>D-28 to D-1 | Eligibility<br>visit <sup>a</sup><br>D-3 to D-1 | Malaria<br>inoculation<br>day<br>D0 | Post-<br>inoculation<br>phone<br>contact<br>D1 to D3 | Malaria<br>monitoring <sup>b</sup><br>D4 to D7 | OZ439 and PQP<br>treatment and<br>clinical unit<br>confinement<br>D8 to D11 | Out-patient<br>monitoring<br>D12 to D42±2 | Rescue<br>treatment<br>with Riamet®<br>D42±2<br>or earlier if<br>required | EOS visit<br>D45±2 |
| Informed consent & BDI | X | | | | | | | | |
| Medical history,eligibility & prior medications | Х | | X | | | | | | |
| Drug & alcohol screen | Х | | X | | | X | | | |
| Full physical examination | Х | | | | | | | | Х |
| Abbreviated physical examination | | | Х | | | Xr | | | |
| Symptomdirected physical examination | | | | | Х | Х | Х | Х | |
| Vital sign assessment | X | | X | | X | X | X | X | Х |
| ECG | Х | | X | | | Χj | | X | Х |
| Urinalysis | X | X | | | | X <sup>k</sup> | X | | Х |
| Haematology & biochemistry | X | X | | | | X | X | X | Х |
| Coagulation profile | X | | | | | | | | |
| G6PD testing | X | | | | | | | | |
| RBC alloantibody | X | | | | | | | | Х |
| Serology | X | | | | | | | | Х |
| Serumβ-hCG pregnancy test | Χď | X | | | | | | | Х |
| Urine β-hCG pregnancy test | | | X | | | X | | | |
| Safety serum storage | | | X | | | | | | X |
| AEs & concomitant medications | | | X | X | Х | X | Х | Х | X |
| Malaria clinical score | | | Х | | X | X | ΧI | Х | X |
| Malaria 18S qPCR blood sampling | | | Х | | Х | X | Xm | Х | Х |
| Parasite lifecycle stage qRTCR blood sampling | | | | | | | Х | Х | Х |
| OZ439 and PQP concentration | | 1 | | | | | ,, | 1/0 | |
| blood sampling | | | | | | X | X | Xs | |
| Phone call or text message | | | | | | | | Xn | |
| Malaria inoculum | | | Xa | | | | | | |
| OZ439 and PQRreatment | | | | | | X | | | |
| Riame® treatment | | | | | | | | Х | |
| Primacin <sup>TM</sup> treatment <sup>i</sup> | | | | | | | | X | |

| Immune cell characterisation (optional) | Χ° | Χ <sup>P</sup> | Χq | Х | Х |
|-------------------------------------------|----|----------------|----|---|---|
| Complement regulatory proteins (optional) | Χ° | | Χq | Х | Х |

PQP: piperaquine phosphateOS: End of StudyBDI: Beck Depression InventoryECG: electrocardiogramG6PD: glucose6-phosphate dehydrogenase, RBC: red blood cell, PK: pharmacokinetic, PD: pharmacodynamic, qPCR: quantitative polymerase chain reaction, qRTPCR: reverse transcription qPCR

- <sup>a</sup> An additional safety visit will occur between Day and Day-1 to collect samples for haematology, biochemistry and urinalysis, unless screening laboratory assessments were conducted within this period.
- <sup>b</sup> Daily visits until qPCR positive, and then twice daily visits u02/2439 and PQP treatment.
- <sup>c</sup> Symptomdirected physical examination will be performed only if clinically indicated at the discretion of the vestigator (see Appendix3 for a list of symptoms and signs of malaria
- <sup>d</sup> Performfollicle stimulating hormone test (pestenopausal females) at screening.
- <sup>e</sup> To be performed at screening visit
- f May be performed at thevestigators discretion, most probably pre and post administration of rescue medidations assure level of gametocytaemia.
- g Cannulate subjects with an indwelling intravenous cannulahtenmalaria inoculum, and record which arm is utilised annulate subjects with an indwelling intravenous cannula for the malaria inoculum, and record which arm is utilised. Administeritate ma inoculum of ~2 800 viable P. falciparum 3D7 infected human RBCs intravenously in the morning (approximately 9:00 AM). Observe for a minimum of 60 minutes after inoculation to evaluate for immediate adverse reactions. Educate subjects on signts anschstymp malaria (Appendix 3). Emphasise to subjects the important returning on the nominated day (approximately Day 8), or as advised by the clinical unit staff, for IMP antimalarial treatment. Provide subjects with diary cards and thermometers to record emarging readings during the study in the event of provides. Subjects will also record symptoms and concomitant medications on the diary cards during the study
- hRiame® treatment will occur on Da∳2±2, or earlierif there is failure of clearance fined asailure to clear parasitaemia by at least 10-fold at 72 hours postMP administration recrudescence of parasitaer (defined as 5 000 blood stage parasites/mL and a 2-fold increase within 48 hours, or a malaria clinical score of the theorem increase within 48 hours.
- i Primacin<sup>TM</sup> treatment if required (Section 6.1.5)
- j ECG to be performed triplicate at 4, 6, 8, 12, 24 and 72 hoursestOZ439 and PQP dosingnd prior to Riamet treatment at the Investigators discretion

<sup>&</sup>lt;sup>k</sup> At the time of **a**lmission to clinical unit only.

<sup>&</sup>lt;sup>1</sup>Only if vital signs are abnormal, or at threvestigators discretion.

<sup>&</sup>lt;sup>m</sup> 18s malariato beperformed Day 12/2am & pm), Day 13(am & pm) then 3x per week until EOSt Investigators discretion

<sup>&</sup>lt;sup>n</sup>Phone call for 3 days to ensure adheren@iaone® treatment

<sup>°</sup> Blood collection prenoculation

<sup>&</sup>lt;sup>p</sup>Blood collection Day 4 visit

<sup>&</sup>lt;sup>q</sup>Blood collectionpre-OZ439 and PQP dosing

<sup>&</sup>lt;sup>r</sup> Abbreviated physical examination OZ439 and PQP dosing

s Blood collection for OZ439 and PQP PK at Day±22lf Riame® treatmentoccurs prior to Day 452 the PK collection will continue as per scheduled timpeoints
#### 7.4 JUSTIFICATION FOR SENSITIVE PROCEDURES

Not applicable.

## 7.5 CONCOMITANT MEDICATIONS, TREATMENTS, ANDPROCEDURES

Concomitant medications, treatments and procedures are those occurring from malaria inoculation until the end of the study (last visit). Those occurring prior to inoculation are classified as prior medications, treatments and procedures. Medications taket in 28 days before the malaria inoculation will be recorded as prior medication. Prior and concomitant medications, treatments and procedures permitted in this study are outlined in the inclusion/exclusion criteria (Section 5.1 and 5.2).

On inoculationday, subjects will be questioned in relation to relevant aspects of compliance with the study protocol, including drug intake since their screening visit. Details of all other drugs taken (prescription and overhe-counter, systemic and topical administra) will be recorded at this time and appropriate action taken. **Three**stigatormay permit the use of ibuprofen up to 1.2 g/day or paracetamol up to 4 g/day, for treatment of headache or other pain if rethuirerofenis the preferred treatment for chadache or pain. To minimise the risk of liver enzyme elevation paracetamol is to be avoided if possible, however paracetamol may be required by some subjects and as such is not a prohibited substantage medication taken from inoculation day to the end of the study (last visit), for treatment of a medical condition and timing of each dose should be recorded.

# 7.5.1 PRECAUTIONARY MEDICATIONS, TREATMENTS, AND PROCEDURES

Not applicable.

#### 7.6 PROHIBITED MEDICATIONS, TREATMENTS, ANDPROCEDURES

Subjects will be informed and reminded of the following restrictions during recruitment, the informed consent process, and during screening and other assessments:

- Subjects should not consume grapefruit or Seville oranges from inoculation day until the end
  of thestudy.
- Subjects should not consume quinine containing foods/beverages such as tonic water, lemon bitter, from inoculation day until the end the Riamet treatment.
- Subjects should not eat any poppy seeds in the 24 hours before the following interest screening, inoculation day, and day of admission for OZ439 and PQP treatment.

- Subjects should not eat or drink any food or beverages that contain alcohol (e.g. beer, wine, and mixed drinks) during confinement at the clinical unit and also 24 hours prior to each alcohol breath test. Subjects should not drink more than 2 standaks pein day from 24 hours before inoculation until the end of the Riantestatment.
- Subjects should not consume beverages that contain xanthine bases (e.g. Red Bull, coffee)
  during confinement at the clinical unit. Subjects should not consume more thamg400
  caffeine per day, equivalent to more than 4 cups of coffee, from inoculation until the end of
  the Riame® treatment.
- Subjects should not use tobacco during confinement at the clinical unit. Subjects should not smoke more than 5 cigarettes or equivalent day from inoculation until the end of the Riamer treatment.

# 7.7 PROPHYLACTIC MEDICATIONS, TREATMENTS, AND PROCEDURES

Not applicable.

#### 7.8 RESCUE MEDICATIONS, TREATMENTS, AND PROŒDURES

The rescue medications used in this study are RametPrimacin<sup>TM</sup> (if required). See details in Section 6.If a subject vomits or cannot tolerate oral drugs, then artesunate will be administered intravenously as described in Section 6.1.5.

#### 7.9 SUBJECT ACCESS TO STDY AGENT AT STUDY CLOSURE

Not applicable.

# 8 ASSESSMENT OF SAFETY

#### 8.1 SPECIFICATION OF SAILTY PARAMETERS

Safety of a single combined dose of OZ439 and PQP will be evaluated by the incidence, severity and relationship of observed and selforted AE's, AESI's and SAE's. Other safety parameters monitored during this study include physical examination, vital signs, clinical biochemistry, haematology, urinalysistriplicate ECG, serology, RBC alloantibody testing, and malaria clinical score. See Sections 7.1 and 7.2 for details of these procedures. All safety parameters will be recorded in the eCRISafety monitoring will be specified in a safety management plan.

## 8.1.1 DEFINITION OF AES (AE)

An AE is defined as any untoward medical occurreince, anyunfavourableand unintended sign (including an abnormal laboratory finding) ymptom or disease that occurs is ubject during the

course of the studyind which does not necessily have a causal relationship with this treatment (i.e., whether not considered drugelated)

A treatmentemergentAE (TEAE) is an event that emerges following treatment with the investigational medicinal products (IMP3Z439 and PQ)P, having been absent pineatment, or worsens relative to the pteeatment state.

#### AEs include but are not limited to

- A new symptom, sign or medical condition.
- A disease or medical condition detected or diagnosed during the course of the study even though it may have been present prior to the start of the study.
- An exacerbation of a prexisting medical condition or disease.
- An increase in frequency or intensity of a poxesting episodic disease or medical condition.
- Continuous persistent diseasesymptoms present at study start that worsen following the start of the study.
- An abnormal assessment (e.g. change on physical examination, ECG findings) if it represents a clinically significant finding that was not present at study start or worsened during the course of the study.
- An abnormal laboratory test result if it represents a clinically significant finding, symptomatic or not, which was not present at study start or worsened during the course of the study or led to dose reduction, interruptionpermanent discontinuation of study treatment.

Borderline abnormal laboratory findings and other objective assessments should NOT be routinely captured and reported as AEs, as they will be collected and analysed separately. However, abnormal laboratory fixings or other objective measurements that meet the following criteria should be captured and reported in the AE section of the eCRF:

- the result meets the criteria for reporting as an SAE
- the test result is associated with accompanying symptoms, and/or
- it requires additional diagnostic testing or medical/surgical intervention, and/or
- it leads to a change in trial dosing, or discontinuation from the trial, significant additional concomitant drug treatment, or other therapy, and/or
- it is considered by then vestigatoror Sponsor to be clinically significant or represent a clinically significant change from baseline.

Merely repeating an abnormal test, in the absence of any of the above conditions, does not constitute an AE. Any abnormal test result that is the ined to be an error does not require reporting as an AE.

Surgical procedures themselves are not AEs; they are therapeutic measures for conditions which may, or may not, be AEs.

Certain information, although not considered an AE, must be recorded, reported, and followed up as indicated for an SAE (see Section 8.4.2 Serious AE Reporting). This includes:

- Pregnancy exposure to an IMP. If a pregnancy is confirmed, use of the IMP must be discontinued immediately. Information about pregnancy exposure includes the entire course of pregnancy and delivery, and perinatal and neonatal outcomes, even if there are no abnormal findings. Both maternal and paternal exposures are considered other reportable information. For exposure involving the female partner of a male subject, the necessary information must be collected from the subject, while respecting the confidentiality of the partner.
- Lactation exposure to an IMP with or without an AE.
- Overdose of an IMP as specified in this protocol with or without an AE.
- Inadvertent or accidental exposure to an IMP with or without an AE

# 8.1.2 DEFINITION OF SERIOUS AES (SAE)

A seriousAE (SAE) is defined as an AE whidalfils at least one of the following criteria:

Results in death.

Is life-threatening

The term "lifethreatening" in the definition of "serious" refers to an event in which the subject was at immediate risk of death at the time of the event; it doesenot r to an event which hypothetically might have caused death if it was more severe.

Requires inpatient hospitalisation or prolongs existing hospitalisation, unless this is for:

- Elective or preplanned treatment or standard monitoring for a-existing condition that is unrelated to the study and has not worsened since the start of the study.
- Cosmetic surgery, or for social reasons, or respite care in the absence of any deterioration in the subject's general condition.

Results in persistent or signification ability/incapacity.

Is a congenital abnormality or birth defect.

Is considered medically important

 Medical and scientific judgement should be exercised in deciding whether other AEs are to be considered serious, such as important medical events threat threat immediately lifethreatening but may jeopardise the subject or may require intervention to prevent one of the other outcomes listed in the definition above. Examples of such events are: intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias; convulsions that do not result in hospitalisation; development of drug dependency or drug abuse.

## Constitutes a possible Hy's Law case

O Hy's Law case is defined as a subject with any value of alanine or aspartate aminotranserasegreater than 3 ULN together with an increase in total bilirubin to a value greater than 2 xULN and not associated to an alkaline phosphatase value greater than 2 xULN (FDA Guidance on Drug Induced Liver Injury: Premarketing Clinical Evaluation[2009]).

A Suspected Unexpected Serious Adverse Reaction (SUSAiR) any SAE where a causal relationship with thenalariainoculum (3D7) or the IMPs QZ439 and PQP is at least a reasonable possibility, and the event is not listed in the (s) and/or Summarof Product Characteristics.

# 8.1.3 DEFINITION OF AES OF SPECIAL INTERES (AESI)

An AESI (serious or nonserious) is one of scientific and medical concern specific to the sponsor's product or programme, for which ongoing monitoring and rapid communication by the Investigator to the sponsor could be propriate Such an event might require the rinvestigation in order to characterise and understand it. Depending on the nature of the event, rapid communication by the trial sponsor to other parties (e.g., regulators) might also be warranted (CIOMS VI, ICH E2F, 2010) Any abnormalities listed be well as AESI:

# Hepatic:

- any ALT or AST above5xULN
- an elevation in bilirubin 2xULN
- any AST or ALT above 2xULN and (TBL > 1.5x ULN or INR > 1.4)
- any AST or ALT above 2xULN with the appearance of fatigue, nawseating, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (eosinophil percent or count above the ULN)

#### Cardiac:

- QTcB or QTcF at any time >480smac,
- bundle branch block (except right bundle branch block that was present prior to IMP administration)
- any arrhythmiaexcept:
  - · sinus bradycardia that is
    - clinically asymptomatic, and
    - not associated with any other relevant ECG abnormalities
  - sinus tachycardia that is
    - clinically asymptomatic, and
    - associated with a body temperature >360 and
    - not associated with any other relevant ECG abnormalities
  - respiratory sinus arrhythmia,

- wandering atrial pacemaker,
- isolated, single premature atrial/ventricular complex (i.e. no bigeminy, trigeminy, couplets, triplets or salvos) that does not occur make once in a particular ECG tracing.

#### Haematological:

- HB drop >2.0 g/dL from baseline prior to inoculation
- Absoluteneutrophil count €00/µl.
- Platelet count ₹5,000 /mm3

#### Dermatological:\*

Clinical signs of possible cutaneous adverse reactions such as:

- dermatitis,
- rash,
- erythematous rash,
- macular rash,
- papular rash,
- maculopapular rash,
- pruritic rash,
- pustular rash,
- vesicular rash
- \* if one of these cutaneous reaction is observed and when feasible, pictures of the lesions should be obtained

#### 8.2 CLASSIFICATION OF ANAE

#### 8.2.1 SEVERITY OF EVENT

In addition to determining whether an AE fulfils the criteria for a SAE or not, the severity of AEs experienced by study subjects will be graded according to the Common Terminology Criteria for AEs v4.03published 14 June 2010 (CTCAE v4.03). This guidance provides a common language to describe levels of severity, to analyse and interpret data, to scale the aggregate AE score, and to articulate the clinical significance of all AEs.

The severity of AEs wilbe graded as follows:

Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.

Grade 2: Moderate; minimal, local or nonvasive intervention indicated; limiting agrepropriate instrumental activities of daily living.

Grade 3: Severe or medically significant but not immediatelythifeatening; hospitalisation or prolongation of hospitalisation indicated; disabling; limiting smaller activities of daily living.

Grade 4: Lifethreatening consequees; urgent intervention indicated.

Grade 5: Death related to AE.

A mild, moderate, or severe AE may or may not be serious (see Section 8.1.2). These terms are used to describe the intensity of a specific event. Medical judgment should be used obya case case basis.

Seriousness, rather than severity assessment, determines the regulatory reporting obligations.

For guidance for assigning severity of the malaria, the purplesigned malaria clinical score will be used (Section 7.1.1).

#### 8.2.2 RELATIONSHIP TO STUDY AGENT

The Investigatorwill decide if AEs are related to any of the study agents or procedures. Where possible, a distinction should be made between events considered related to the malaria challenge agent the IMPs rescue treatments of other protocol-mandated procedures. The assessment of causality will be made using the following definitions:

#### Unrelated

This category is applicable to those AEs which are judged to be clearly and incontrovertibly due to extraneous causes (disease, environment, etc.) and do not meet the criteria for the relationship listed under unlikely, possible or probable.

#### Unlikely

In general, this category is applicable to an AE which meets the following criteria (must have the first two):

- 1. It doesnot follow a reasonable temporal sequence from administration of any of the study agents.
- 2. It may readily have been produced the subject's clinical state, environment or toxic factors, or other modes of therapy administered to the subject.
- 3. It does not follow a known pattern of response to the study agents.
- 4. It does not reappear or worsen when any of the study agentsædnenineistered.

#### Possible

This category applies to those AEs in which the connection with any of the study agents appears unlikely but cannot be ruled out with certainty. An AE may be considered possible if or when (must have the first two):

- 1. It follows a reasonable temporal sequence from administration of any of the study agents.
- 2. It may have been produced by the subject's clinical state, environment or toxic factors, or other modes of therapy administered to the subject.
- 3. It follows a known pattern of respse to any of the study agents.

#### Probable

This category applies to those AEs which are considered, with a high degree of certainty, to be related to the study agents. An AE may be considered probable if (must have the first three):

- 1. It follows a reasondb temporal sequence from administration of any of the study agents.
- It cannot be reasonably explained by the known characteristics of the subject's clinical state, environment or toxic factors, or other modes of therapy administered to the subject.
- It disappears or decreases on cessation or reduction in dose.
- 4. It follows a known pattern of response to any of the study agents.
- 5. It reappears on **redministration**.

#### 8.2.3 EXPECTEDNESS

An AE is regarded as a manexpected everify its nature or severity is notionsistent with the applicable reference safety information of approved manufacturer's prescribing information for marketed drugs). Events that add significant information on the specificity, severity or frequency of previously described reactions, also regarded as unexpected.

Expected AEs from the malaria infection listed in Appendix and the for the 3D7 inoculum [35]. Expected AEs from the antimalarial drugs used are listed **10746** 91B [38] and the EMA European Public Assessment Reptot PQP, Riame Consumer Medicine Information, Primacin Consumer Medicine Information, and artesunate WD Public Assessment Report 2011 (see Appedix 1).

# 8.3 TIME PERIOD AND FREQUENCY FOR EVENT ASSISSMENT AND FOLLOW-UP

All AEs must be documented and followed up by Ithæstigatoruntil:

- the event is resolved, or
- no further medically relevant information in relation to the event can be expected, and
- the Investigator considers it justifiable to terminate the followp.

Events that are unresolved at the time of the subject's last follow-up visit should continue to be followed up by thenvestigatorfor as long as medically indicated. The Sponsor retains the right to request additional information for any subject with ongoing AE(s)/SAE(s) at the end of the study, if judged necessary.

All AEs should be treated appropriate. The Investigator will decide upon the appropriate action to be taken in response to an AE, which may include one or more of the following:

- No action taken (i.e. further observation only).
- Dosing with the IMP is withheld and the subject withdrawn from the study.
- Administration of a concomitant medication.
- Hospitalisation or prolongation of current hospitalisation (event to be reported as an SAE).
- Other.

In a case of occurrence of SAEs, regardless of whether or not it is judged to be claudent guerantimalarial drugelated, the subject will receive appropriate care under clinical supervision until all the symptoms of the SAEs have diminished or resolved and the subject's condition improved.

For ongoing AEs, care will be provided for **aripel** of time as specified in the clinical site work instruction protocols. However, if the nature of the ongoing AE is determined **byvetest**igator as not being inoculumor antimalarial drugassociated, the subject will be advised to visit his/her own general practitioner for further clinical care that he might require.

#### 8.4 REPORTING PROCEDURES

#### 8.4.1 AE REPORTING

It is the Investigator's responsibility to document and report all AEs occurring in the study whether spontaneously reported by the subject, observed by Inthrestigator (either directly or by laboratory or other assessments), or elicited by general questioning. The pebisdroftion for collection of AEs extends from the time of inoculation up to the end of the study; these AEs must be recorded as pages of the eCREvents reported prior to this will be recorded as medical history, unless the symptoms worse indutthe study.

The following information should be recorded for all AEs:

- Description of the AE.
- Dates and times of onset and resolution of the event.
- Duration of the event in hours.
- The time of onset relative timoculum, or the OZ439 and PQP treatmemntd/or the antimalarial rescue drugs
- Seriousness of the AE (SAE or not).
- Severity of the event.
- Action taken in response to the event (including treatment required).
- Outcome of the event.
- Relationship of the event to the study agents or procedures (causality assessment), including inoculum, IMPs, rescue medication, or any other treatment or procedure conducted during the study.
- Changes in the severity of an AE will be documented to alkowessment of the duration of the event at each level of severity.
- AEs worsening in severity will be considered unresolved and those reducing in severity will be considered resolving.
- AEs characterised as intermittent requilibrecumentation of onset and dration at each episode.
- Only one AE is reported if there is a variation in intensity (with highest intensity for final CSR Tables): the description will also report the various severities over time,
- If the AE resolves and then reoccur at a later date: the AE are reported
- All malaria-specific AEs will be tabulated and results graded according to a purpose designed malaria clinical score table (Section 7.1.1).

8.4.2 SERIOUSAE REPORTING

The Investigatorwill take immediate appropriate action in response to SAEs to ensure subject safety and in an attempt to identify the causes of the eventln vestigatorwill notify Prime Vigilance, of any SAE within 24 hours of becoming aware of the event. The notifion should be in writing by email or fax, and documented on a standard SAE reporting form.

## SeriousAE Reporting:

Prime Vigilance

Email: MMV@primevigilance.com

Fax: +44 800 471 5694

Medical Director
Stephan Chalon, MD, PhD
Medicines for Malaria/enture
Route de PreBois 20
1215 Geneva 15
Switzerland

Email: chalons@mmv.orRepresentative

#### Medical Monitor

Dr. med Michael Marx MD

Medical Director

ICON Clinical Research Internal Tel: 7123 1568

ExternalTel: +49 6103 904 1568 Mobile: (+49) 172 677 7401

Email:STUDY-MA-DL-3037-0010Blinded@iconplc.com

The Investigatorwill complete a followup SAE report within 14 days of the SAE, unless no further information is available in which case the follow report will be provided soon as new information becomes available. The follow SAE report will be sent to the recipients the initial report as described abo@ther supporting documents may be requested by these parties and will be provided by the requested by the reques

Any SAE that meets the criteria of a SUSAR (Section 8.1.2) will be reported to the TGA by the local sponsor CNS in accordance with the Sponsor's reporting procedures.

#### 8.4.3 UNANTICIPATED PROBLEM REPORTING

Not applicable.

# 8.4.4 AES OF SPECIAL INTERES (AESI)

All AESIs, including those that do not meet the definition of an SAE, must be notified to the Pharmacovigilance provider (Prime vigilance) within 24 hours of the estigator becoming aware of the occurrence of the AE\$ he notification should be in writing by email or fax (Prime vigilance contact details mentioned above in 8.4.2 section) and documented on a standard AESI reporting form. Within 1 business day of receipt of any safety reports (initial or follow reports), Prime vigilance will notify the medical monitor (with the Sponsor medical monitor in copy), the sponsor and the BT of the event and its follows and will include all available information.

The notification of followup information will follow the same procedure and timelines as the initial report.

#### 8.4.5 REPORTING OF PREGNANY

Pregnancyin a female subject on a male subject's female partner during the study should be reported and followed as described beneath. Pregnancy does not constate to and the pregnancy outcome will not be recorded in the eCRF unless it is considered to the an

The Investigatormust notifyPrimeVigilance, in an expedited mannef any pregnancy occurring from the date of informed consent signature consent signature consents after administration consents and PQP. The same process as described for AEs and AESI as designated ion 8.4.2 should be followed. In all cases, the pregnancy mutest followed until birth of the child, and the outcome of the pregnancy and birth reported as above by completing appropriate section of the Pregnancy Report Form used for the initial notification. The timelines of the outcome reporting vary as follows:

- Normal outcomes should be reported within 45 days of birth/delivery
- Abnormal outcomes should be reported in an expedited manner as described in Section8.4.2.

An additional SAE Report form must be completed if the subject or subject's partner sustains a serious eventA ParentChild/Foetus Report (PCFR) must be completed echild/foetussustain an event.

#### 8.5 STUDY HALTING RULES

See Section 5.5.

#### 8.6 SAFETY OVERSIGHT

Safety oversight will be undertaken by the Princilpred estigator and the Medical Monitor who will serve as an independent expert to advise on clinical safety specifically in the situation where expert external advice is required regarding the need for administration of alternative/rescue antimalarial treatment in the circumstance defeatimal response.

The SDRT will be responsible for decisions related to the safety of subjects and the continuation of the study. The role and composition of the SDRT is outlined in the study specific DSRT Charter. The SDRT will be composed of the Princip Investigator Medical Monitor, and a physician with expertise in clinical trials or infectious diseases. TDRS will review the clinical and laboratory safety data as well as the recorded AEs and SAEs. TDRET Snakes recommendations to the Sponsor. These recommendations are approved by tDRTS Chair who signs a letter of recommendation that is sent to the Princip Restigator and the Sponsor.

A review by the SPRT of data from each cohort will be conducted prior to dosing the subsequent cohort. Safety and tolerability data up to Da\$42±2, and PK/PDanalysis outcomes (based on PD data up to Da\$42±2 and PK data up to Da\$45±2) from all subjects who received eatment with OZ439 and PQRvill be required for the reviewA similar analysis will be done at the end of cohort 2 combining cohort and 2 data to decide the d(ss) to be tested in cohort 3 his will be decided by the funding sponsor and Rhiencipal Investigator following review of the data by the SDRT and scientific evaluation.

Additionally, the SDRT may meet to assess any events that trigger the stopping rules or as needed to provide a recommendation and findings to QIMR Berghofer HREC and the Principal Investigator in accordance with the approve DBT Charter.

Whether at a scheduled or unscheduled meeting, **DR**TSwill consider safety signals to determine whether or not they can recommend that the study continue.

The SDRT will also review the safety and tolerability to from the study after completion of the last cohort.

# 9 CLINI CAL MONITORING

It will be the Sponsor's responsibility to ensure that the study is monitored in accordance with the requirements of GCP. The conduct of the study will be reviewed internally eboylinical unit (Q Pharm) in accordance with their standard procedures and work instructions, and GCP guidelines. The study will be monitored according to the SQPtshe monitoring CRO appointed this task by the Sponsoand all protocol deviations will be reported to the Sponsor. Protocol deviations that impacts ubject safety or data integrit will also be reported to the QIMR Berghofer HREC.

During the study, appointed study monitor((sx)) behalf of the Sponsor) will visit the site to check completeness of subject records, accuracy of eCRF entries, adherence to the protocol and to GCP, progress of enrolment, and to ensure that study agents were stored, dispensed, and accounted for according to specifications. Key study personnel are required to be be assist the study monitor during these visits.

The Investigatorwill be required to give the monitor access to all relevant source documents to confirm their consistency with the eCRF entries. The Spowistorequire full verification for the presence of informed consent, adherence to the inclusion/exclusion criteria, documentation of SAEs, and the recording of data that is used for all primary and safety variables. Additional checks of the consistency of the source data with the eCRFs will be performed according to the study specific monitoring plan. No information in source documents about the identity of the subjects will be disclosed.

## 10 STATISTICAL CONSIDER ATIONS

#### 10.1 STATISTICAL ANALYSIS PLAN

The following sections describe the statistical analysis as it is foreseen when the study is being planned. A detailed Statistical Analysis Plan (SAP) will be finalised and approved prior to database lock and will provide details of all analyses to be **perf**ed as well as the format of listings and tables to be provided for completion of the Clinical Study Report (CSR). Any deviations from the SAP will be described and justified in the final CSR.

For the safety primary endpoint, we hypothesise that indeglatith ~2800 viableP. falciparum 3D7 parasitenfected RBCs and treating with OZ439 and PQP on trial Day 8 will be safe and will result in no SAE, sandwill not cause severe malaria symptoms.

This study is not powered to compare IMP dostest rather to answer the primary objectives.

#### 10.2 ANALYSIS DATASETS

The safety analysis dataset will include all subjects who receive the malaria inoculum. This population will be used to analyse all safety data as well as demographic and baseline data.

The populatio(s) used for analysis of PK, Pand PK/PD analysis ill be defined in the SAP.

## 10.3 DESCRIPTION OF STATSTICAL METHODS

#### 10.3.1 GENERAL APPROACH

This is an adaptive lose finding study using the IBSM model to characterise the K/PD relationship between OZ439 and PQP for the treatment of election.

Continuous data will be summarised using descriptive statistics (mean and standard deviation, or median and interquartile range). Categorical data will besented using the number N() and percentage%) (using the number of subjects without missing data in the calculation).

# 10.3.2ANALYSIS OF THE PRIMARY EFFICACY ENDPOINT(S)

A model-based analysis is foreseton characterise the PK/PD relationship between QZ439 and PQP plasma concentrations and blood stage asexual parasitaemia. For assessing the contribution of each compound and their interaction effect, data of this combination therapy study, will be pooled with data from previous human challenge monotherapy studies for each compound, i.e. QP12C01 (OZ439) and QP13C05 (Piperaquine).

The final PK/PD model will describe time courses of plasma concentrations and of the parasite countsby a nonlinear mixed effets (NLME) modelling approachThe change in parasite count will be modelled as the joint effects of parasite growth and drug concentration

The model will be developed in step wise manner. First, a joint PK model for OZ439 and piperaquine will be establised potentially taking PK drugtrug interaction into account. Second, the PD model will be developed using individual PK parameters as regressors. The effect of each compound on parasite clearance is described by a sigmoidant Edel or related models at take into account time delays of the drug action if appropribe interactions between OZ439 and PQP will be described using the Genter D Interaction (GPDI) model PD interaction scenarios to be tested with the GLDI model include a change in each sdEC50, Emax or EC50 and Enax caused by the other drug.

Graphical displays will be given, where appropriate. Details of the modelling analysis will be described in the modelling analysis plan (MAP).

# 10.3.3ANALYSIS OF THE SECONDARY ENDPOINT(S)

The secondary endpoints are PD and PK parameters.

# PK parameters

Estimation of OZ439 and PQP PK parameters over 28 days afternoin istration of single doses using noncompartmental methods:

The following pharmacokinetic parameters will be determined good noncompartmental method from plasma concentration data from all cohort  $\Delta UC_{0-168h}$ ,  $AUC_{last}$ ,  $AUC_{0-inf}$ ,  $C_{max}$ ,  $t_{max}$ ,  $t_{1/2}$ ,  $t_{lag}$ ,  $C_{168h}$ , CL/F, Vz/F and  $\lambda_{inf}$ . These data will be summarized descriptively by treatment and dose.

For calculation of descriptive statistics of blood concentrations, values below the LLOQ will be set to zero.

Pharmacokinetic parameters will be determined gSTATA® (version14.0 or highe)r.

# PD parameters

Parasite Reduction Ratio (PRR). The PRR of asexual parasites will be based on the decay of parasitaemia after drug treatment determined by malaria 18S qmeRRR for asexual parasites will be estimated using the slope of the optimal fit of theliogar relationship of the parasitation decay[45]. The optimal fit can be derived using summarised replicate parasitaemia data, which have been cleaned by dealing with potential outliers, values below the limit of detection and non detectable values (ND). The optimal fit of the kingear parasitaemia by-time relationship is determined by using left and right censoring to systematically remove the potential lag phase and tail phase of the parasitaemia decay. The decay rate, estimated slopth coefficient from the log-linear decay regression of qPCR data, will be calculated for each subject. The overall cohort dose specific PRR will be estimated with its 95% CI by calculating the weighted average slope estimate and corresponding standardor (SE) using an inverseariance method. Only subjects who have optimal regression models with appropriate fit contribute toward the places for PRR. Details are presented in the SAP.

Parasite clearance halflife (t 1/2). The Pt 1/2 will be derived from the optimal decay rate. Details regarding the calculation will be in the SAP.

Percentage of subjects with recrudescence of parasitaemia percentage of subjects with recrudescence parasitaemia parasitaemia tollowing treatment with OZ439 and PQIPhis will be determined by the number of subjects who experience rudescence which defined as \$\geq 5000\$ blood stage parasites/mL and a-fold parasitaemia increase within 48 hours, onceurrence of malaria symptoms with a malaria clinical score > This will be determined by parasite lifecycle qRT PCR.

#### 10.3.4SAFETY ANALYSES

The overall number and percentage of subjects with at least one AE (and SAE) will be tabulated over the entire study period. All AE data will be summarisephooled treatment group and study period, i.e. Day 0 to Day 8 (inoculum), Day 8 after dosing or earlier to Day (12Z439 and PQP) and Day 12±2 after dosing (Rescue treatment) to (EOS visit).

Treatment emergent AE's will also be summarised with frequency counts by MedDRA system organ class (SOC; i.e. body system) and preferred term (PT), for each pooled treatment group and by Study period.

Vital signs, routine safety laboratory data and ECG parameters will discented in data listing and will be summaised descriptively by treatment group and by protocol specified tiproxint.

Where applicable both absolute values and change from baseline (inoculation) IMPs administration) will be presented and listings of clinically relevant abnormal laboratory transfer be generated.

The safety and tolerability of a single combined dose of OZ439 and PQP will be evaluated by the incidence, severity and relationship of observed and septified AEsup to trial Day 422.

# 10.3.5 ADHERENCE AND RETENTION ANALYSES

Not applicable.

#### 10.3.6 BASELINE DESCRIPTIVESTATISTICS

Demographic data will be summarised by descriptive statistics and will include total number of observations (n), mean, standard deviation (SD) and range for continuous variables and number and percentages with characteristics for dichotomous variables.

The subject disposition will be summarised. Study completion, study withdrawals, exclusions and violations will be summarised and the reasons for withdrawal, exclusions and violations will be listed.

Medical history, current medical conditions, previous **and**comitant medications, results of laboratory screening tests, drug and alcohol screening tests and any other relevant baseline information will be listed by subject and cohort.

#### 10.3.7 PLANNED INTERIM ANALYSES

#### 10.3.7.1 SAFETY REVIEW

A review of the safety and tolerability data from the preceding cohort will be conducted by the SDRT prior to inoculation of the next cohoAtll safety and tolerability at up to and including Day 35±2will be required for each review.

See Sectin 5.5 for study stopping rules.

#### 10.37.2 EFFICACY AND PK REVIEW

A review of the parasitaemia datand PK data analysis from the preceding cohort will be conducted by the LSRT prior to inoculation of the next cohort. All data up to and including Day 42±2 will be required for each review review of the PK/PD analysis based on PD data up to Day 42±2 and PK data up to Day 5±2 postdose from the preceding cohort(s) will be conducted by the SDRT prior to inoculation of the next cohort.

#### 10.3.8 ADDITIONAL SUB-GROUP ANALYSES

Not applicable.

#### 10.3.9MULTIPLE COMPARISONMULTIPLICITY

Not applicable.

#### 10.3.10 TABULATION OF INDIVI DUAL RESPONSE DATA

All individual subject data will be listed by measure and time point.

#### 10.3.11 EXPLORATORY ANALYSES

No formal statistical analyses are planned for exploratory endpoints.

#### 10.4 SAMPLE SIZE

A total of up to 24 healthy subjects will be enrolled in the study (to 3 cohorts of 8 subjects each). Subjects will be malaria naïve healthy male or female adults, aged betweeners old, who meet all of the inclusion criteria and none of the exclusion criteria.

In each cohort, if more than 2 discontinuations due to sate ty related reasons occur; additional subjects may be recruited to replace the discontinued subjects on agreement with the study sponsor.

Historically, 8 participants in a dose has proven to be sufficient to characterise the effect of a drug on malariaparasite kinetics following induction of IBSM of healthy subjects.

#### 10.5 MEASURES TO MINIMIZE BIAS

#### 10.5.1ENROLLMENT/ RANDOMIZATION/ MASKING PROCEDURES

Randomisation will be performed r subjects in all cohorts. The 8 subjects f all cohorts will be randomised to one of the dose groups each cohort (see Table 1 and 2 Section 4.) after inoculation day but prior to Day. 8

The randomisation schedule will be generated by a statistician using a validated Aystepyn. of the randomisation schedule will be sent to the clinical unit pharmacistiaircal unit project manager.

#### 10.5.2EVALUATION OF SUCCESS OF BLINDING

Not applicable.

# 10.5.3BREAKING THE STUDY BLIND/SUBJECT CODE

Not applicable.

# 11 SOURCE DOCUMENTS AND ACCESS TO SOURCE DATA/DOCUMENTS

The Investigatorwill maintain source documents for each subject in the study. Information entered into eCRFs will be traceable to these source documents in the subject's filevestigatormust certify that the datæntered into the eCRFs are complete and accurate. After database lock, the Investigatorwill retain copies of the subject data for archiving at the investigational site.

Upon request, then vestigato(s)/institution(s) will permit direct access to soudzeta/documents for trial-related monitoring, audits, Ethics Committee review, and regulatory inspection(s) by the Sponsor (or their appropriately qualified delegate) and Regulatory Authorities. Direct access includes examination, analysis, verification are production of records and reports that are important to the evaluation of the trial.

# 12 QUALITY ASSURANCE AN D QUALITY CONTROL

Data management, including the development and management of a secure database, will be performed in accordance with regulatorequirementsCNS will review the data entered into the eCRFs by clinical unit staff for completeness and accuracy. A formal querying process will be followed whereby the data management team will request the clinical site staff to clarify any apparent eroneous entries or inconsistencies and will request additional information from the clinical site as required.

Medical history/current medical conditions dAEs will be coded using the Medical dictionary for regulatory activities (MedDRA) terminology (weign 20.1 or higher). Prior and concomitant medications are to be coded using the WHO-DDE dictionary (March 2014 or later).

After all data have been captured and reviewed, all queries have been resolved with the site and any protocol noncompliances that we identified during the data management processes have been confirmed by the site, the database will be declared to be complete and accurate, it will be locked and made available for data analysis. Any changes to the database after that time may only bemade by the data manager, in consultation with the Sponsor and in accordance with documented database unlock and relock procedures.

Clinical monitoring will be conducted as described in Section 9.

Audits may be carried out by Sponsor quality assurances septatives, local authorities or authorities to whom information on this study has been submitted. All documents pertinent to this study must be made available for such inspections after adequate notice of intention to audit.

#### 13 ETHICS/PROTECTION OF HUMAN SUBJECTS

#### 13.1 ETHICAL STANDARD

The study will be conducted in accordance with the protocol approved by the QIMR Berghofer HREC, the principles of the Declaration of Helsinki (Recommendations guiding Medical Doctors in Biomedical Research Involving Human Participants, Fortaleza, Br@2B)2 the NHMRC National Statement on Ethical Conduct in Human Research (2007, updated May420)25)d the Note for Guidance on Good Clinical Practice Annotated with TGA Comments (CPMP/ICH/135/95), as adopted byethoustralian Therapeutic Goods Administrationally 2000) [47].

The Investigatorwill minimise any discomfort experienced by subjects during the study. The only invasive procedures will be the intravenous inoculation of the malaria inoculum and the blood collection by cannulation/venepunœurThe maximum amount of blood be collected from an individual in the study would be up to approximates mL (Appendix 2)

| Blood Volume | Time-frame | mL (approximately) |
|---------------------|---------------------------|--------------------|
| Main study | Screening to Day 30 | 239 |
| Optional components | Screening to Day 30 | 173 |
| Total | Screening to Day 30 | 412 |
| Main study | Screening to Day 45 (EOS) | 297 |
| Optional components | Screening to Day 45 (EOS) | 201 |
| Total | Screening to Day 45 (EOS) | 497 |

The total volume of blood drawn from each subject will not exceed 450 mL in any 30 weeking period. This volume includes allowance for unscheduled safety and qPCR assessments that may be required at the discretion of the Princilpred estigator the Sponsor to ensure subject safety.

#### 13.2 ETHICAL REVIEW

The protocol Participant Information Sheets and informed consent forms will be reviewed by the QIMR Berghofer HREC, and no study activities will be initiated prior to approval from the Berghofer HREC. All amendments and addenda to the protocol and consent forms will similarly be submitted to the QIMR Berghofer HREC for approval prior to their implementation.

Changes to the final study protocol can only be made with the prior consent of the Principal Investigator the Sponsor and the IMR BerghoferHREC. All such changes must battached to, or incorporated into, the final protocol, and communicated to all relevant member battached to, staff and, if appropriate, to study subjects. All deviations from this study protocol will be included in the trial master file and included in the SR. An assessment of the significance of each protocol deviation will be given in the CSR. All deviations/amendments will be reported to Sponsor and the QIMR Berghofer Project Manager. The different types of amendments are discussed below.

#### Non-substantibamendment

Administrative or logistical minor changes require a -substantial amendment. Such changes include but are not limited to changes in study staff or contact details (e.g., Sponsor instead of CRO monitors) or minor changes in the packagingabelling of study drug. An amendment deemed to be negubstantial must have no ethical implications.

The implementation of a negrubstantial amendment may be done without notification to the QIMR BerghoferHREC. It does not require their approval or too stigned by then vestigator The QIMR BerghoferHREC will be notified of these negrubstantial changes in the next submission round, with the annual study report or study close out reposite ever will be submitterized to QIMR BerghoferHREC.

#### Substantial amendment

Significant changes require a substantial amendment. Significant changes include but are not limited to: new data affecting the safety of subjects, change of the objectives/endpoints of the study, eligibility criteria, dose regimestudy assessments/procedures, treatment or study duration, with or without the need to modify the Participant Information Sheet and Informed Consent.

Substantial amendments are to be approved both BerghoferHREC. The implementation of a substantial mendment can only occur after formal approval by the BerghoferHREC and must be signed by the vestigator

# <u>Urgent amendment</u>

An urgent amendment might become necessary to preserve the safety of the subjects included in the study. The requirements rfapproval should in no way prevent any immediate action being

taken by thenvestigator the Sponsor in the best interests of the subjects. Therefore, if deemed necessary, almovestigator implement an immediate change to the protocol for safetynesa. This means that, exceptionally, the implementation of urgent amendments will occur before submission to and approval by toleral Berghofer HREC.

In such cases, then vestigator must notify the Sponsor within 24 hours. A related substantial amendment will be written within 10 working days and submitted to the IR Berghofer HREC, together with a description of the steps that have already been taken in regard to implementation of this amendment.

# HREC approval of future research

In the event that ther Procipal Investigator the Sponsor want to perform testing on the samples that is not described in the protocol, additio QdMR BerghoferHREC approval will be sought. This may be done if a subject has consented to blood storage for use in future (Section 13.3.1)

#### 13.3 INFORMED CONSENT PRŒESS

# 13.3.1CONSENT/ASSENT AND OTHER INFORMATIONAL DOCUMENTS PROVIDED TO SUBJECTS

The Participant Information Sheet and informed Consent Form describes in detail the study agents, study procedures, and risks. Subjects will also receive an Informed Consent for Blood Storage and an option to grant permission to be contacted about futurdly involvement.

Details regarding the optional study components will be provided in a separate Participant Information Sheet and subjects agreeing to participate in these components will provide specific written consent for this Subjects will also receive an Informed Consent for Blood Storage and an option to grant permission to be contacted about future study involve Regusal to participate in the optional study components will not jeopardise a subjects' participation in the main study.

Subjects will also receive the product insert for artesunate, and the Consumer Medicine Information for Riamet and Primacin (if required; Appendix 1). Subjects may also receive the Consumer Medicine Information for any other registered antimalarial agents irretitation these are required.

#### 13.3.2CONSENT PROCEDURES NO DOCUMENTATION

During the initial screening visit/recruitment, potential subjects will read the Participant Information Sheet. Then vestigator clinical unit staff will explain the study via the Participant Information Sheet and the potential subjects will be encouraged to ask questions. Individuals

willing to be considered for inclusion in the study will sign and date the informed Consent Form in the presence of anvestigator Subjects will be given a copy of their signed informed Consent Form. Once the subject has consented to the study, the precautic screening activities may commence. See Section 7.3.1 for further details.

#### 13.4 SUBJECT AND DATA CONFIDENTIALITY

Subjects will beinformed that their data will be held on file by Parm and that these data may be viewed by staff of Pharm (including, where necessary, staff Parm other than the named Investigatos).

Upon request, then vestigato(s)/institution(s) will permitdirect access to data and documents for trial-related monitoring, audits, Ethics Committee review, and regulatory inspection(s) by the Sponsor (or their appropriately qualified delegates) and Regulatory Authorities (see Section 11).

Subjects will also benformed that a report of the study will be submitted to the Sponsor and may also be submitted to government agencies and perhaps for publication, but that they will only be identified in such reports by their study identification number, and their gemetage. The Investigatorundertakes to hold all personal information in confidence.

Subjects will be informed that samples collected for the purposes described in the protocol will be sent to Sponsor's nominated national or international laboratory for assessment.

### 13.4.1RESEARCH USE OF STORD HUMAN SAMPLES, SPECIMENSOR DATA

Samples and data collected during this study will be used to achieve the study objectives.

Samples and data will be stored according that m and QIMR Berghofer SOPs, and access will be limited to authorised personnel. Biological samples will be retained for the time required to complete analysis, and may then be discarded.

#### 13.5 FUTURE USE OFSTORED SPECIMENS

As part of the study, safety serum samples will be stored indefinitely Pana (2011) Pana (2011) As part of the study, safety assessments that may later be indicate; etc consent to this storage and the use of the sample for safety assessments, when they sign the informed Consent Form for the study.

For all other samples, consent must be obtained from the subjects to store and use their samples for future research. Consentwill be obtained via the Informed Consent for Blood Storage that subjects receive during recruitment/screening. Subjects can decide if they want their samples to be

used for future research or have their samples destroyed at the EOS. A subject's decision can be changed at any time prior to the EOS by notifying the study doctors or nurses in writing. However, if a subject has consented to future use and some of their blood has already been used for research purposes, the information from that **eas**ch may still be used.

Any future research using the stored samples that is beyond the current study will be reviewed by the QIMR Berghofer HREC (Section 13.2). All samples will be stored at QIMR Berghofer in accordance with the laboratory SOPs. Threestigatorwill ensure that confidentiality will be maintained continuously in all future research that involves use of these samples. The vials containing the samples of the consented subjects will be coded and the identifying information will not be released to any unauthorised third party. The subjects can also choose (via the Informed Consent for Blood Storage Form) for the samples to the beddelled with only the study number, malaria strain and visit. No genetic testing will be performed on the starredless without obtaining consent from the subjects. The stored samples will not be sold or used directly for production of any commercial product. There are no benefits to subjects in the collection, storage and subsequent research use of their samplesorts eabout future research done with subject samples will NOT be kept in their health records, but a subject's samples may be kept with the study records or in other secure areas.

## 14 DATA HANDLING AND RE CORD KEEPING

#### 14.1 DATA COLLECTION AND MANAGEMENT RESPONSIBILITIES

Each subject will have a clinical file (source data) and case report form (CRF, for protocol specific data) into which relevant data will be recorded. All recording will be done only in black ink. Corrections will only be made by drawingsingle line through the incorrect entry, writing the correction in the nearest practicable space, initialling and dating the correction. Correction fluids are not allowed.

A log of names, signatures and initials of all staff authorised to enter data into a subject's Clinic File and CRF will be kept. Upon completion of each study visit, all CRFs will be reviewed internally by the clinic for omissions or apparent errors so these can be corrected without delay. Any corrections made after the review and signature of the Principal internal and will required reauthorisation (electronic sign off) by the Principal Investigator

#### 14.2 STUDY RECORDS RETENTION

All source data, clinical records and laboratory data relating to the study will be retained in the archive of the clinical unit(Q-Pharm) for a minimum of 15 years after the completion of the study. Data will be available for retrospective view or audit by arrangement with the Chief Executive

Officer of the clinical unit. Written agreement from the Sponsor must precede destruction of the same.

#### 14.3 PROTOCOL DEVIATIONS

Protocol Deviation: protocol deviation is any departure or chargen, and addition to, the study design or procedures defined in the protocol that has received approval by the competent authorities and favourable opinion from the ethics committees.

Important Protocol Deviation: an important protocol deviation (sometiefierred to as a violation) is a protocol deviation that has or has the potential to affect the rights, safety-or well being of the trial subjects and may impact the integrity (completeness, accuracy and reliability) of the data to a degree that the data of usable.

NTF: a noteto file is a record that documents in detail actions taken, important decisions made or explains a sequence of events where no other detailed record exists to enable the conduct of the trial to be reconstructed.

All protocol deviations will be documented in the trial master file and included in the CSR. An assessment of the significance of each protocol deviation will be discussed in the CSR.

All NTFs, protocol deviations and important protocol deviations are to be viewed by interpal Investigator delegate (QIMRBerghoferProjectManager) and signed by the recipal Investigator

All NTFs, protocol deviations and important protocol deviationils assessed and significance assigned at the end of each cohort by the SDRT.team

All, important protocol deviations ill be reported by the clinical site to the Sponsor and the Sponsors request the QIMR Berghofer HRE@s early as possible, builthin 7 days. A protocol violation report form provided by QIMR Berghofer will besed for this purpose

All protocol deviations will be reportedly the clinical site the QIMR Berghofer PMas early as possible but within 7 days and to the Sponsorat the end of each cohora. protocol deviation report form provided by QIMR Berghoferill be used for this purpose

Protocol deviation logswill be submitted by the clinical site the Sponsor and QIMR Berghofer HREC via inclusion with the annual report.

#### 14.4 PUBLICATION AND DATA SHARING POLICY

The data management, statistical and mæddwriting team appointed by the Sponsor will collaborate to provide a detailed CSR upon conclusion of the study. This will include appendices of all tables and listings generated during the analyses of data. The tables and listings will be

provided by CNS. The Sponsor undertakes to ensure that all safety observations made during the conduct of the trial are documented in this report.

Publication and reporting of results and outcomes of this trial will be accurate and honest, undertaken with integrity and insparency and in accordance with the relevant clauses outlined in the QIMR Berghofer Policy on Criteria for Authors [148]. QIMR Berghofer and the Principal Investigator have a responsibility to ensure that results of scientific interest arising from the clinical trials are appropriately published and disseminated. Publication of results will be subjected to fair peerreview. Authorship will be given to all persons pidding significant input into the conception, design, and execution or reporting of the research according to the QIMR Berghofer Policy on Criteria of Authorship. No person who is an author, consistent with this definition, will be excluded as an author known known the hard permission in writing. Authorship will be discussed between researchers prior to study commencement (or as soon as possible thereafter) and reviewed whenever there are changes in participation. Acknowledgment will be given to collaborating institutions and hospitals and other individuals and organisations providing finance or facilities. All conflicts arising from disputes about authorship will be reviewed by the QIMR Berghofer Director.

In any press releases, publications or presentations, MMV's financial contribution to the study and its participation in the collaboration shall be expressly acknowled@tMR Berghofer agrees that MMV will be entitled to access all the-identified clirical trial data upon completion of the trial. Data will not be released publicly until the manuscript is accepted for publication. In the case of no publication, information will only be released to the public and media in accordance with the QIMR BerghofeCorporate Media Strategy Poli[M9]. However, thenvestigatorundertakes not to make any publication or release pertaining to the study and/or results of the study without the Sponser's prior written consent, being understood that the Sponsor will not unreasonably withhold its approvalThe Sponsor has the right to publish the results of the study at any time.

The Investigatorshall not use the name(s) of the Sponsor and/or of intropers in advertising or promotional material or publication without the prior written consent of the Sponsor. The Sponsor shall not use the name(s) of the setigator and/or the collaborators in advertising or promotional material or publication without aving received his/her and/or their prior written consent(s).

MMV or the local sponsowill ensure that the key design elements of this protocol are posted in a publicly accessible database such as Australian New Zealand Clinical Trials Registry (ANZCTR) or Clinicaltrials.gov. In addition, upon study completion and finalisation of the study,represent results of this trial will be either submitted for publication in an open access journal and/or posted in a publicly accessible database of clinical tries ults.

# 15 STUDY ADMINISTRATION

#### 15.1 STUDY LEADERSHIP

See Section 1 for key roles.

#### 15.2 LIABILITY/INDEMNITY/ INSURANCE

The study Sponsor will ensure sufficient insurance is available to enable it to indemnify and hold the Investigato(s) and relevant staff as well as any hospital, institution, Ethics Committee or the like, harmless from any claims for damages for unexpected injuries, including death, that may be caused by the subject's participation in the study but only to the extent that the claim is not caused by the fault or negligence of the subjects revestigato(s). The Sponsor adheres to the guidelines of Medicines Australia for injury resulting from participation in a company sponsored trial, including the provision of 'No-fault clinical trial insurance'.

# 16 CONFLICT OF INTEREST POLICY

No conflicts of interest are applicable in this study.

# 17 LITERATURE REFERENCE S

- 1. WHO, 2017.
- 2. Dondorp, A.M., et al. Artemisinin resistance in Plasmodium falciparumalaria. New England Journal of Medicine, 200361(5): p. 455-467.
- 3. Woodrow, C.J. and N.J. White he clinical impact of artemisinin resistance in Southeast Asia and the potential for future spreateMS Microbiol Rev, 201741(1): p. 3448.
- 4. Straimer J., et al. Drug resistance. K1-propeller mutations confer artemisinin resistance in Plasmodium falciparum clinical isolate science, 2015347(6220): p. 4281.
- 5. Burrows, J.N., et al. New developments in antialarial target candidate and product profiles. Malar J, 2017.16(1): p. 26.
- 6. Phyo, A.P., et al., Antimalarial activity of artefenomel (OZ439), a novel synthetic antimalarial endoperoxide, in patients with Plasmodium falciparum and Plasmodium vivax malaria: an operhabel phase 2 trial Lancet Infect Dis, 2016.16(1): p. 6169.
- 7. McCarthy, J.S., et al Linking Murine and Human Plasmodium falciparum Challenge Models in a Translational Path for Antimalarial Drug Development imicrob Agents Chemother, 201660(6): p. 366975.

- 8. Macintyre, F., et al.A randomised, doublelind clinical phase II trial of the efficacy, safety, tolerability and pharmacokinetics of a single dose combination treatment with artefenomel and piperaquine in adults and children with uncomplicated Plasmodiu falciparum malaria. BMC Med, 2017.15(1): p. 181.
- 9. ANZCTR Trial ID: ACTRN12611001203943An experimental study to characterize molecular signatures during early Plasmodium falciparum blood stage infection in healthy male volunteers2011.
- 10. ANZCTR Trial ID: ACTRN12612000323820\( \text{An experimental study to characterize the effectiveness of Lariam (Registered Trademark Mefloquine) against early Plasmodium falciparum blood stage infection in healthy volunteers 2012.
- 11. ANZCTR Trial ID: ACTRN12612000814875 experimental study to characterize the effectiveness of OZ439 against early Plasmodium falciparum blood stage infection in healthy volunteers 2012.
- 12. ANZCTR Trial ID: ACTRN12613000533796 and Phase I/Ib study to investigate the safety, tolerabilityand pharmacokinetic profile of DSM265 in healthy subjects and to assess the antimalarial activity of DSM265 in healthy subjects with an induced blood stage Plasmodium falciparum infectio@013.
- 13. ANZCTR Trial ID: ACTRN12613000565741An experimental stdy to characterize the effectiveness of piperaquine against early Plasmodium falciparum blood stage infection in healthy volunteers2013.
- 14. ANZCTR Trial ID: ACTRN12613000698774 in experimental study to characterize the effectiveness of griseofulvinæigst early Plasmodium falciparum blood stage infection in healthy volunteers 2013.
- 15. ANZCTR Trial ID: ACTRN12613001040752 experimental study to characterize the effectiveness of ferroquine against early Plasmodium falciparum blood stage infection i healthy volunteers 2013.
- 16. ANZCTR Trial ID: ACTRN12614000781640 an Adproof of concept study to assess the effect of ACT451840 against early Plasmodium falciparum blood stage infection in healthy subjects2014.
- 17. Bijker, E.M., et al., Protection against malaria after immunization by chloroquine prophylaxis and sporozoites is mediated by preerythrocytic imm@nitog.Natl Acad Sci U S A, 2013.110(19): p. 78627.
- 18. Cheng, Q., et al Measurement of Plasmodium falciparum growth rates in vivostacte malaria vaccines Am J Trop Med Hyg, 199757(4): p. 495500.
- 19. ClinicalTrials.gov ID: NCT02281344A proof-of-concept study to assess the effect of MMV390048 against early Plasmodium falciparum blood stage infection in healthy participants 2014.

- 20. ClinicalTrials.gov ID: NCT02389348A proof-of-concept study to assess the effect of a range of doses of combined therapy with OZ439 and DSM265 against early Plasmodium falciparum blood stage infection in healthy participarate15.
- 21. ClinicalTrials.gov ID: NCT02543086A phase 1 interventional sequential single site study to characterize the effectiveness of oral KAE609 in reducing asexual & sexualstateged P. falciparum following inoculation in healthy volunteers & subsequent infectivity to mosquitoes 2015.
- 22. Duncan, C.J., et allimpact on malaria parasite multiplication rates in infected volunteers of the proteinin-adjuvant vaccine AMAC1/Alhydrogel+CPG 7909PLoS One, 2011. 6(7): p. e22271.
- 23. Lawrence, G., et al. Effect of vaccination ith 3 recombinant asexustage malaria antigens on initial growth rates of Plasmodium falciparum in-immune volunteers. Vaccine, 200018(18): p. 192531.
- 24. McCarthy, J.S., et al.A pilot randomised trial of induced bloodage Plasmodium falciparuminfections in healthy volunteers for testing efficacy of new antimalarial drugs. PLoS One, 20116(8): p. e21914.
- 25. Payne, R.O., et alpemonstration of the bloostage Plasmodium falciparum controlled human malaria infection model to assess efficatethe P. falciparum apical membrane antigen 1 Vaccine, FMP2.1/ASQI Infect Dis, 2016.
- 26. Pombo, D.J., et allmmunity to malaria after administration of ultraw doses of red cells infected with Plasmodium falciparurbancet, 2002360(9333): p. 616617.
- 27. Sanderson, F., et allood-stage challenge for malaria vaccine efficacy trials: a pilot study with discussion of safety and potential value of J Trop Med Hyg, 2008.8(6): p. 87883.
- 28. ClinicalTrials.gov ID: NCT02431637Blood stage challengetudy to assess mosquito transmissibility in participants inoculated with Plasmodium falcipar2015.
- 29. ClinicalTrials.gov ID: NCT02431650 proof-of-concept study to assess the effectiveness of OZ439 as a gametocytocidal and transmission blocking taige experimental P. falciparum infection 2015.
- 30. ClinicalTrials.gov ID: NCT02573857A phase Ib study to characterise the antimalarial and transmission blocking activity of a single dose of DSM265 or OZ439 in healthy subjects with induced blood sta@smodium falciparum or Plasmodium vivax infection 2015.
- 31. Krause, A., et al.Pharmacokinetic/pharmacodynamic modelling of the antimalarial effect of Actelion451840 in an induced blood stage malaria study in healthy subpartsClin Pharmacol, 203.

- 32. McCarthy, J.S., et al. Efficacy of OZ439 (artefenomel) against early Plasmodium falciparum bloodstage malaria infection in healthy volunteed Antimicrob Chemother, 2016.
- 33. McCarthy, J.S., et al.A. Phase II pilot trial to evaluate safety aetficacy of ferroquine against early Plasmodium falciparum in an induced bletage malaria infection study. Malar J, 2016:15: p. 469.
- 34. Pasay, C.J., et a P. iperaquine Monotherapy of Drugusceptible Plasmodium falciparum Infection Results in Rapidle arance of Parasitemia but Is Followed by the Appearance of Gametocytemia Infect Dis, 2016214(1): p. 10513.
- 35. Investigators BrochureBlood stage Plasmodium falciparum challenge inoculum P. falciparum 3D7 (BSPC) v8.0 e2017, QIMR BerghofeMedical Research Institute.
- 36. Warrell, D.A., Essential malariology4 ed ed. 2002, London: Arnold.
- 37. S, C., et al. Poster presentation: Moderate and severe LFT elevations in controlled human P. falciparum malaria infection model: recent experience atiture review and mechanistic hypotheses American Society of Tropical Medicine and Hygiene: 65th Annual Meeting 2016.
- 38. Investigators Brochure: Medicines for Malaria Vent@**Z**439 (artefenomel) Version 12.0 21 December 201**Z**017, Medicines fo**M**alaria Venture.
- 39. Myint, H.Y., et al., Efficacy and safety of dihydroartemisirpirperaquine. Trans R Soc Trop Med Hyg, 2007101(9): p. 85866.
- 40. Ratcliff, A., et al., Two fixeddose artemisinin combinations for drugsistant falciparum and vivax maria in Papua, Indonesia: an opdabel randomised comparisolancet, 2007.369(9563): p. 75765.
- 41. Karunajeewa, H., et al.Şafety evaluation of fixed combination piperaquine plus dihydroartemisinin (Artekin) in Cambodian children and adults with miala J Clin Pharmacol, 200457(1): p. 939.
- 42. Mytton, O.T., et al., Electrocardiographic safety evaluation of dihydroartemisinin piperaquine in the treatment of uncomplicated falciparum malania. J Trop Med Hyg, 2007.77(3): p. 44750.
- 43. European Medicines Agency Eurartesim: European Public Assessment Reportoduct Information. Updated 2016.
- 44. Australian Therapeutic Goods Administrationaccess to unapproved therapeutic goods: Clinical trials in Australia 2004.
- 45. Marquart, L., et al., Evaluating the pharmacodynamic effect of antimalarial drugs in clinical trials by quantitative PCRAntimicrob Agents Chemother, 20159(7): p. 4249 59.

- 46. National Health and Medical Research Countriational statement on ethical conduct in human researct 20072007. p. 1-95.
- 47. Australian Therapeutic Goods Administration for Guidance on Good Clinical Practice (GCP) (CPMP/ICH/135/952000.
- 48. QIMR Berghofer Medical Research Instituteolicy on the criteria for authorship2008.
- 49. QIMR Berghofe Medical Research Instituted edia relations policy2010.

# **APPENDIX**

Appendix 1: Product information and consumer medicine information

# Riame®

- Product Information (TGA, updated August 2016)
- Consumer Medicine Information (TGA, updated Decen20215)

# Primacin<sup>TM</sup>

- Product Information (TGA, updated February 2017)
- Consumer Medicine Information (TGA, updated February 2017)

#### Artesunate

• WHO Public Assessment Report (2011)

Appendix 2: Total blood volume

| Procedure | Sample | Volume per<br>sample<br>(mL) | No. samples per subject | Total volume per subject (mL) |
|---|---|---|---|---|
| | Haematology | 2 | 7 | 14 |
| | (including<br>G6PD) | 4 | 2 | 8 |
| | Biochemistry<br>/biomarker(may | 5 | 6 | 30 |
| Laboratory<br>Safety | include<br>Serology CRP, | 8.5 | 3 | 25.5 |
| Assessment | Coagulation profile | 2.7 | 1 | 2.7 |
| | Safetyserum<br>storage | 5 | 2 | 10 |
| | RBC alloantibody | 4 | 2 | 8 |
| Bioanalysis | PK analysis | 4 | 21 | 84 |
| Cannulation | Discard | 2 | 19 | 38 |
| Malaria<br>Monitoring | Malaria 18S<br>qPCR | 2 | 36 | 72 |
| | Parasite<br>lifecycle stage<br>qRT-PCR | 2 | 2 | 4 |
| Main study total (mL) | | | | ~297 |
| | ImmuneCell | 53 | 2 | 106 |
| Exploratory<br>(optional) | Characterisation | 26 | 3 | 78 |
| | Complement<br>Regulatory<br>Proteins | 2 | 8 | 16 |
| Additional optional exploratory totathL) | | | ~203 | |
| Main study and exploratory components(mL) | | | ~497 | |

This table is indicative and may vary based on qPCR levels and safety-toplosamples. Additional blood samples may be taken for unscheduled safety and qPCR assessments as required by the Investigator provided the total volume taken during the studysdoct exceed 450 mL during any period of 30 consecutive days.

# Appendix 3: Symptoms and signs of malaria

Following challenge via the intravenous malaria parasite inoculation and during the plustige period, the following signs and symptoms of malaria be monitored:

# Signs of malaria

- Fever (oral temperature of  $\geq 38^{\circ}$ C)
- Chills/shivering/rigors
- Tachycardia
- Hypotension

# Symptoms of malaria

- Headache
- Myalgia (muscle ache)
- Arthralgia (joint ache)
- Fatigue/lethargy
- Malaise (general discomfort/uneasiness)
- Sweating/hot spells
- Anorexia
- Nausea
- Vomiting
- Abdominal discomfort

# Appendix 4: Beck Depression Inventory

# Appendix 5: Version History

| Version | Date | Author(s)/Reviewer(s) | Revisions |
|---------|---------|-----------------------|-----------------------------|
| 1.0-1.1 | 29.1.18 | Rebecca Webster | Minor typographical updates |
| 1.1-2.0 | 19.3.18 | Rebecca Webster | See table below |
| 2.0-3.0 | 30.4.18 | Rebecca Webster | See table below |
| 3.0-4.0 | 20.8.18 | Rebecca Webster | See table below |

# Summary of Changes to QP17C16Version 1.1 to 2.0)

| Protocol Section(s) | Change | Rationale |
|---|---|---|
| Abbreviations | <ul> <li>Added 2additional<br/>abbreviations</li> </ul> | Missing from initial protocol |
| Protocol Summary<br>and Objectives and<br>Purpose | Added optional exploratory objectives and endpoints | Additional scientific exploratory objectives have been added to the protocol These are optional studie and participants that choos to participate will sign a separate consent form |
| Key Roles | <ul> <li>An additional independent<br/>medical monitor has been<br/>added to the trial key roles</li> <li>Data management, site<br/>monitoring and regulatory<br/>function personnel has been<br/>added to the trial key roles</li> </ul> | <ul> <li>The sponsor requested an additional medical monitor</li> <li>A specific person from the local sponsor has been identified to perform this role</li> </ul> |
| 4.1 | Added additional text<br>regarding the exploratory<br>study components | Additional scientific exploratory objectives have been added to the protocol These are optional studies and participants that choos to participate will sign a separate consent form |
| 6.1.1 | Change of sucrose provider<br>from MMV to Q-Pharm | <ul> <li>Updated to highlight that<br/>sucrose will be provided by<br/>the phase 1 site pharmacy</li> </ul> |
| 7.1.1 | <ul> <li>Added additional text to further explain;</li> </ul> | Clarification and completeness of protocol |

| 7.2.2 | <ul> <li>ECG procedural requirement</li> <li>exploratory study blood sampling</li> <li>medical diary cards and temperature selfecording</li> <li>Added details about;</li> <li>PK blood collection and processing</li> <li>optional exploratory components</li> <li>optional exploratory components</li> </ul> | Clarification and completeness of protocol and updated information regarding theadditional exploratory objectives |
|---|---|---|
| 7.3 Study Schedule | <ul> <li>Added blood collection for optional exploratory components at each relevan time-point</li> <li>Added a subject diary card check at all relevant time points</li> </ul> | Updated with information<br>related to the additional<br>exploratory objectives |
| 7.3.7 | Updated schedule of events | Clarification of schedule of<br>participant activities in line<br>with above described text |
| 13.1 | Updated study total blood<br>volume to include explorator<br>components blood volume | Updated with information related to the additional exploratory objectives |
| 14.3 | <ul> <li>Added text about reporting or protocol deviations and violations</li> </ul> | Clarification of reporting obligations |
| Appendix 2 | Updated total blood volume | Updated due to additional<br>blood volume being<br>requiredfor exploratory<br>optional components |

# Summary of Changes to QP17C1(Version 2.0 to 3.0)

| Protocol | Change | Rationale |
|---|---|---|
| Section(s) Protocol Summary, 4.1, 6.1.5 7.3.3 | Added criteria for IMP administration (malaria clinical score >6) and definition of recrudescence a a criterion for rescue medication administration (defined as ≥5 000 blood stage parasites/mL and a 2 fold increase within 48 hours or a malaria clinical score >6 | was deemed necessary<br>rather than just a defined<br>time-point for these<br>activities |
| Key Roles | <ul> <li>An additional coinvestigator<br/>has been added to the trial k<br/>roles</li> </ul> | |
| 2.3 IMP<br>risks | <ul> <li>Added vasovagal, orthostation<br/>hypotension and atrial<br/>fibrillation to the risks section</li> </ul> | identified |
| 5.1<br>Inclusion<br>criteria | <ul> <li>Change from 50 to 40 mmHg ≤ diastolic blood pressure</li> <li>Added male subjects with female partners that are surgically sterile, or male subjects who have undergon sterilisation and have had testing to confirm the succes of the sterilisation may also be included.</li> </ul> | |
| 5.2<br>Exclusion<br>criteria | <ul> <li>Change Participation in any investigational product study within the 12 weeks precedir the study to Participation in any investigational product study within the 12 weeks preceding IMP administration.</li> <li>Clarification that Symptomatimostural hypotension at screening, irrespective of the decrease blood pressure, or asymptomatic postural</li> </ul> | |

| | <ul> <li>hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 2-3 minutes when changing from supine to standing position, could be peated if abnormal</li> <li>Clarification and separation of severe allergic reaction, anaphylaxis and convulsions</li> </ul> | |
|---|---|---|
| 7.1.1 | Stated that the mean of the<br>three ECGs would be<br>recorded | Clarification of protocol |
| 7.2.1 | <ul><li>Added MCV to haematology</li><li>Added coagulation testing</li></ul> | Missed in previous protoco |
| 7.3.2 | <ul> <li>Updated schedule of events</li> <li>CRP will be included in all biochemistry except screening</li> <li>Urine for urinalysis will be collected at EOS</li> <li>Coagulation added to table of events</li> </ul> | |
| 7.3.3 | An additional malaria PCR time point added | <ul> <li>Required to collect blood<br/>for PRR every 6 hours afte<br/>initial administration of<br/>IMP</li> </ul> |
| 8.1.3 | <ul> <li>Changed ALT or AST above<br/>3x ULN to 5x ULN</li> <li>QTcB or QTcF prolongation<br/>from baseline claffication of<br/>parameter</li> <li>Clarification of<br/>haematological AESI</li> </ul> | Clarification and specification of appropriate AESI's for malaria challenge studies |
| 13.1<br>Appendix 2 | Updated blood volume | Updated since added coagulation profile |

# Summary of Changes to QP17C1@Version 3.0 to 4.0)

| Protocol<br>Section(s) | Change | Rationale |
|---|---|---|
| Protocol<br>Summary,<br>4.1, | Added planned dose regime<br>for Cohort 2 post SDRT<br>meeting and scientific data<br>evaluation | Cohort 2 doses selected after SDRT review. |
| Protocol<br>Summary,<br>4.1,<br>7.3.3<br>8.6,<br>10.3 | Updated trial day naming convention | Study Day numbers were updated as per studgesign schemænd study flowchart for consistency. |
| 7.3.3 | Added ECG assessment to<br>time of rescue treatment<br>administration | Provide additional safety data prior to rescue treatment |
| 5.2 | Updated citrus consumption<br>till the EOS rather than end of<br>Riamet treatment | |
| 7.6 | <ul> <li>Updated alcohol grams into<br/>units and standard drinks<br/>(Australian)</li> </ul> | Updated to be consistent with the eCRF |
| 8.4.5 | Updated pregnancy wording | WOCBP can be included in<br>this studyas per inclusion<br>criteria under the condition<br>of usage of highly effective<br>method ofbirth controland<br>therefore this section<br>needed to be revised |
| 10.5 | Changed randomisation to occur afterinoculation but prior to Day 8. | Logistically this provides<br>more time for the clinical<br>site to prepartor dosing. |
| 7.1.1 | Added on study IBSM specific ranges or ECGs and vital signs | Provide additional information and alignment with eCRFguidelines |
| 7.3.2<br>7.3.3 | Changed symptom directed physical examination to a compulsory abbreviated | Provide additional safety assessment opfarticipants |

| | physical examinatio <b>p</b> rior to inoculum and drug dosing | prior to inoculum and drug dosing |
|---|---|---|
| 7.3.3 | Added text regarding assessments to be performer if participants are administered antimalarial rescue treatment prior the (Day 42) scheduled time point. | To ensure safety assessments which are required to be performed at the end of rescue treatmen are captured in the protoco if participants are provided antimalarial rescue therapy prior to the scheduled time point. |
| 7.2.1<br>7.3 | Defined CRP as a biomarker | <ul> <li>CRP is a biomarker and no<br/>a biochemistry safety<br/>assessment</li> </ul> |
| 7.2.2<br>7.3.3 | <ul> <li>Added the following wording<br/>to applicable protocolsections<br/>"Malaria monitoring will<br/>continue until a minimum of<br/>one negative 18S qPCR is<br/>detected post rescue therapy</li> </ul> | number of negative qPCR required after rescue therapy to consider a subject successfully rescued |
| 7.3.4 | <ul> <li>Changed capturing anarial<br/>clinical score to benandatory<br/>at EOS</li> </ul> | To provide additional safety information |
| 7.3.7 | <ul> <li>Updated SoE table</li> <li>Added abbreviated physical exa</li> <li>Added rescue treatment column</li> </ul> | • |